#### **Quotient Confidential**



Doc No: DOC-181160 Version: 0.13 Status: Ready for Approval

Doc Name: QSC300553 Reporting and Analysis Plan NCT #: NCT06612255

Project Number: QSC300553

## **REPORTING AND ANALYSIS PLAN**

A Phase 1, Single Part, Partially Randomised, Open-Label Study to Evaluate the Relative Bioavailability of a Taste-Masked Delafloxacin Powder of Oral Suspension with Oral Delafloxacin Tablet Reference in Healthy Subjects

Quotient Study Number: QSC300553

Sponsor Study Number: ML-DEL-101-3727-1

Melinta Subsidiary Corporation

Sponsor: A Wholly Owned Subsidiary of Melinta

Therapeutics, LLC 389 Interpace Parkway, Parsippany, NJ 07054 US

Date of RAP: 24 Jun 2024

Status of RAP: Final v1.0

#### SPONSOR/QUOTIENT SCIENCES CONFIDENTIAL

This Reporting and Analysis Plan may not be reproduced or communicated to a third party without the written permission of Melinta Therapeutics, LLC (Melinta).

# Quotient Sciences

#### **Quotient Confidential**

Doc No: DOC-181160 Version: 0.13 Status: Ready for Approval

Doc Name: QSC300553 Reporting and Analysis Plan

Project Number: QSC300553

## **Document Version History**

| Version<br>Number | Reason for Update | Updates Made | Updated By: | Date |
|---|---|---|---|---|
| v1.0 | Finalisation of v1.0 | NA | | 24 Jun 2024 |

| Author | |
|-----------------------------------------------------|------|
| See electronic signature at the end of the document | Date |
| (Quotient) | Date |
| Approvers | |
| See electronic signature at the end of the document | |
| (Quotient) | Date |
| (Maclinto) | Date |
| (Melinta) | |
| | Data |
| (Melinta) | Date |

 $\boxtimes$ Tick here if this document will be following an electronic approval route in Veeva. Signatures will be found on an accompanying page.

| 1 | | i abie of | Contents | |
|---|---|---|---|---|
| 1 | | | Table of Contents | 4 |
| 2 | | | List of Abbreviations | 7 |
| 3 | | | Introduction | . 10 |
| | 3.1 | | Responsibilities | . 10 |
| | 3.2 | | Definitions. | . 10 |
| | | 3.2.1 | Subject Definitions | |
| | | 3.2.2 | Definition of Treatments | |
| | | 3.2.3 | Definition of Visits | . 11 |
| 4 | | | Objectives and Endpoints | . 12 |
| 5 | | | Study Design | . 12 |
| | 5.1 | | Brief Description | . 12 |
| | 5.2 | | Criteria for In-Study Decisions | . 14 |
| | | 5.2.1 | Decision Points | |
| | 5.3 | 5.2.2 | Criteria for Dose Level and Prandial Status Selection | |
| | 5.4 | | Randomisation (including Replacement Subjects) | |
| | 5.5 | | Blinding Issues | |
| 6 | | | Populations and Analysis Sets | |
| U | | | | |
| | 6.1 | | Safety Population and Safety Analysis Set | |
| | 6.2 | | Pharmacokinetic Population and Pharmacokinetic Analysis Set(s). | . 16 |
| | 6.3 | | Taste/Palatability Population and Taste/Palatability Analysis Set(s) | 16 |
| 7 | | | Subject Disposition, Demographics and Baseline Characteristics | . 17 |
| | 7.1 | | Screening Failures | . 17 |
| | 7.2 | | Subject Disposition and Withdrawals | . 17 |
| | 7.3 | | Analysis Populations | . 17 |
| | 7.4 | | Analysis Sets and Subsets | . 18 |
| | 7.5 | | Demographic Characteristics and Lifestyle Details | . 18 |
| | 7.6 | | Medical/Surgical History | . 18 |
| | 7.7 | | Prior and Concomitant Medication | . 18 |
| | 7.8 | | Other Baseline Characteristics | . 19 |
| 8 | | | Efficacy | . 19 |
| 9 | | | Pharmacokinetics | . 19 |
| | 9.1 | | Plasma PK Parameter Estimation | . 19 |

| 9.2 | 9.1.1<br>9.1.2<br>9.1.3 | Definition of Plasma PK Parameters | 21 |
|---|---|---|---|
| 9.3 | | Concentration and PK Figures | |
| 9.4 | | Concentration and PK Listings | |
| 9.5 | | Statistical Analysis of PK Parameters | |
| 0.0 | 9.5.1 | Relative Bioavailability | |
| | 9.5.2 | Food Effect and Optional Dose Proportionality | 25 |
| 9.6 | 9.5.3 | Statistical Figures for Analysis of Pharmacokinetic Data Interim PK Analysis | |
| 10 | | Taste Assessments | |
| 10.1 | | Summary Tables for Taste Assessments | |
| 10.2 | | Listings for Taste Assessment | 27 |
| 11 | | Safety Assessments | 27 |
| 11.1 | | Extent of Exposure and Treatment Compliance | 27 |
| 11.2 | | Meal Details | 27 |
| 11.3 | | Adverse Events | 27 |
| | 11.3.1 | Summary Tables for Adverse Events | |
| 11.4 | 11.3.2 | Listings for Adverse Events | |
| 11.4 | 11.4.1 | Summary Tables for Laboratory Evaluations | |
| | 11.4.1 | Listings for Laboratory Evaluations | |
| 11.5 | | Vital Signs | |
| | 11.5.1 | Summary Tables for Vital Signs | |
| 11.6 | 11.5.2 | Listings for Vital Signs | |
| 11.0 | 11.6.1 | Summary Tables for ECGs | |
| | 11.6.2 | Listings for ECGs | 33 |
| 11.7 | | Physical Examination | 34 |
| 12 | | Interim Statistical Analyses | 34 |
| 13 | | Changes in the Conduct of the Study or Planned Analysis | 34 |
| 13.1 | | Changes in the Conduct of the Study | 34 |
| 13.2 | | Changes to the Planned Analyses | 34 |
| 13.3 | | Any Other Relevant Changes | 34 |
| 14 | | Overall Considerations | 34 |
| 14.1 | | Statistical Programming and Analysis | 34 |
| 14.2 | | Quality Control of Summary Tables, Figures and Listing | |
| Statis | stical Ana | alysis | |

| | 14.2.1 | Quality Control - Summary Tables | 37 |
|---|---|---|---|
| | 14.2.2 | Quality Control - Figures | 37 |
| | 14.2.3 | Quality Control - Data Listings | |
| | 14.2.4 | Quality Control - Statistical Analysis | 38 |
| 15 | | SAS Data Transfer | 38 |
| 16 | | Programming Conventions | 38 |
| 17 | | Reference List | 38 |
| 18 | | Index of Tables | 40 |
| 19 | | Index of Figures | 43 |
| 20 | | Index of Listings | 45 |
| 21 | | Mock Tables | 48 |
| 22 | | Mock Figures | 73 |
| 23 | | Mock Listing | 81 |
| Append | ix 1: Sch | nedule of Assessments | 110 |
| Append | ix 2 <sup>.</sup> Exa | mple Taste/Palatability Questionnaire | 112 |

#### 2 List of Abbreviations

ADaM analysis data model

ADR adverse drug reaction

AE adverse event

ATC anatomical therapeutic chemical

AUC area under the curve

BLQ below the limit of quantification

BMI body mass index

BP blood pressure

CDISC Clinical Data Interchange Standards Consortium

CHMP Committee for Medicinal Products for Human Use

CI confidence interval

CS clinically significant

CSR clinical study report

CV% coefficient of variation

CVw% intra-subject variability

D 'substantial' decrease from baseline for vital signs parameters

DP decimal place

ECG electrocardiogram

eCRF electronic case report form

Frel relative bioavailability

GMR geometric mean ratio

h hour

H flag used for value that is above normal reference range

HR heart rate

'substantial' increase from baseline for vital signs parameters /

I

increase in QTcF interval from baseline

ICH International Council for Harmonisation

IMP investigational medicinal product

ISF Investigator Site File

L flag used for value that is below normal reference range

LLOQ lower limit of quantification

LOD limit of detection

Max maximum

MedDRA Medical Dictionary for Regulatory Activities

Min minimum

n number of subjects with an observation

N number of subjects in the dataset

NA not applicable

NC not calculated

NCS not clinically significant

NR not reportable/no result

NS no sample

PI principal investigator

PK pharmacokinetic

PT preferred term

QC quality control

QTcF QT interval corrected for heart rate using Fridericia's correction

RAP reporting and analysis plan

SAC safety advisory committee

SAE serious adverse event

SD standard deviation

SDTM study data tabulation model

SF significant figure

SI substantial increase in QTcF interval from baseline

SOC system organ class

SOP standard operating procedure

TEAE treatment-emergent adverse event

TFL tables, figures and data listings

WHO World Health Organisation

Abbreviations used for pharmacokinetic parameters and associated flags are defined in Section 9.1.1.

#### 3 Introduction

This document details the following for Quotient Sciences (Quotient) Study QSC300553 (ML-DEL-101-3727-1):

- Criteria to be used for the definition of the populations and analysis sets relating to safety, pharmacokinetic (PK), and taste/palatability data
- Handling of missing data
- Proposed tables, figures, and data listings (TFLs) for demographic, dosing, PK, safety, and taste/palatability data
- Methods for PK parameter estimation and formal statistical analysis

This document has been compiled according to the Quotient standard operating procedure (SOP) "Production of Reporting and Analysis Plans" and has been written based on information contained in the final study protocol (v1.0) dated 19 Mar 2024.

#### 3.1 Responsibilities

The Data Sciences Department at Quotient will be responsible for the production of the following items using Quotient SOPs: Clinical Data Interchange Standards Consortium (CDISC) study data tabulation model (SDTM) and analysis data model (ADaM) datasets, PK parameter estimation and output, and safety and taste/palatability output; including all TFLs, and formal statistical analysis; and the clinical study report (CSR).

Quotient will provide two sets of TFLs during the study:

- Post database lock TFLs (draft) for Melinta review
- Post-review TFLs (final) for inclusion into the CSR

Quotient will be responsible for the quality control (QC) of all deliverables prior to the client review (Section 14.2).

#### 3.2 Definitions

#### 3.2.1 Subject Definitions

An enrolled subject is defined as a subject who signed the informed consent, qualified per the inclusion/exclusion criteria, and was randomised.

#### 3.2.2 Definition of Treatments

Throughout the reporting of the study, investigational medicinal product (IMP) will be referred to as regimen and will be reported as detailed in Table 1 below:

**Table 1 Study Treatments** 

| Period | Regimen | Investigational<br>Medicinal<br>Product | Dose | Route of Administration | TFL Label |
|---|---|---|---|---|---|
| | Α | delafloxacin Tablet (reference) | 450 mg | Oral, Fasted | 450 MG TAB FASTED |
| 1 and 2 | В | delafloxacin Powder for Oral Suspension, reconstituted with orange flavoured vehicle | 450 mg | Oral, Fasted | 450 MG POS FASTED |
| 3 | С | delafloxacin Powder for Oral Suspension, reconstituted with orange flavoured vehicle | 450 mg<br>or<br>XX mg | Oral, Fed<br>or<br>Oral, Fasted | XX MG POS <status></status> |
| 4<br>(optional) | D | delafloxacin Powder for Oral Suspension, reconstituted with orange flavoured vehicle | XX mg<br>or<br>YY mg | Oral, Fed<br>or<br>Oral, Fasted | XX MG POS <status></status> |

The order in which regimens are dosed may be subject to change due to logistical reasons TAB = Tablet, POS = Powder

#### 3.2.3 Definition of Visits

For clinical data, visits will be referred to as Day throughout this document and will be referred to as screening, Day -1 (admission) and Day 1 through to Day 3 and follow-up phone call Day  $6 \pm 1$ . Time points within these days are detailed in the schedule of assessments in Appendix 1.

Baseline is defined as nominally the last measurement recorded prior to dosing of IMP for each study period.

## 4 Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary To determine the relative bioavailability of delafloxacin Powder for Oral Suspension compared to that of oral delafloxacin Tablet reference | Results of the formal statistical analysis of overall exposure (AUC) for delafloxacin Powder for Oral Suspension, compared to oral delafloxacin Tablet reference |
| Secondary To determine the PK of delafloxacin Powder for Oral Suspension formulation | PK parameters for delafloxacin: Tlag, Tmax, Cmax, AUC(0-24), AUC(0-last), AUC(0-inf), lambda-z, Frel,T1/2, CL/F, Vz/F, and MRT, as applicable |
| To determine the relative bioavailability of delafloxacin Powder for Oral Suspension in the fed and fasted state | Results of the formal statistical analysis of overall exposure (AUC) for delafloxacin Powder for Oral Suspension in the fed state compared to the fasted state |
| To provide additional safety and tolerability information for orally administered delafloxacin | Assessment of AEs, vital signs, ECGs, physical examinations, and clinical laboratory tests |
| Exploratory To evaluate the taste/palatability attributes (smell, sweetness, bitterness, flavour, mouthfeel/texture, grittiness, and aftertaste) and overall acceptability of delafloxacin Powder for Oral Suspension | Results of the taste questionnaire |

## 5 Study Design

#### 5.1 Brief Description

This is a Phase 1, single-centre, single-part, partially randomised, open-label, relative bioavailability study in healthy subjects.

It is planned to enrol approximately 16 healthy male and healthy non-pregnant, non-lactating female subjects.

The study will follow the design in Figure 1.

Subjects will undergo preliminary screening procedures for the study at the screening visit (Day -28 to Day -2).

#### Periods 1 and 2

Subjects will be admitted in the morning on the day before dosing (Day -1) in Period 1. Subjects will receive a snack in the evening, after which they will fast overnight from all food and drink (except water) for a minimum of 10 hours. Subjects will be administered IMP on the morning of Day 1 in the fasted state. Subjects will complete a written taste/palatability questionnaire individually and privately following IMP administration (Regimen B only).

Subjects will be randomised in a 1:1 ratio to one of two sequences (AB or BA) immediately prior to dosing in Period 1, for allocation of regimens across Periods 1 and 2.

Blood and urine samples will be collected at regular intervals for PK and safety analysis, as applicable, from admission until 48 hours post-dose during each period. Subjects will remain resident in the clinical unit during the washout period (minimum 4 days) between Periods 1 and 2. Subjects will be discharged from the clinical unit at 48 hours post-dose (Day 3) in Period 2.

Following dosing of Regimens A and B (end of Period 2), there will be an interim decision meeting to review available PK and safety data to decide the dose level and prandial state for Regimen C (Period 3). The Investigator and Sponsor will decide whether to continue to evaluate a 450 mg dose level of delafloxacin Powder for Oral Suspension following a high-fat breakfast, or to evaluate an alternative dose level in the fasted state.

#### Period 3

Subjects will be admitted in the evening on the day before dosing (Day -1). Subjects will fast overnight from all food and drink (except water) for a minimum of 10 hours, and will be administered IMP on the morning of Day 1 in the fasted state (if a different dose level is selected), or approximately 30 minutes after a high-fat breakfast (if a change to prandial state is selected). Subjects will complete a written taste/palatability questionnaire individually and privately following IMP administration.

Blood and urine samples will be collected at regular intervals for PK and safety analyses, as applicable, from admission until 48 hours post-dose (Day 3), at which time subjects will be discharged from the clinical unit.

Following dosing of Regimen C, there will be an interim decision meeting to review available PK and safety data, to decide whether to proceed with optional Period 4 or whether to end the study. If it is decided to end the study, a follow-up phone call will take place on Day  $6 \pm 1$  to ensure the ongoing wellbeing of subjects. If a subject reports any AEs that present a cause for concern, they will be required to attend the clinical unit for an (unscheduled) follow-up visit. End of study is defined as completion of the last follow-up phone call or unscheduled follow-up visit. If it is decided to proceed with optional Period 4, the dose level and prandial state for Regimen D will be determined; the Investigator and Sponsor will decide whether to continue to evaluate the dose level selected for Regimen C following a high-fat breakfast, or to evaluate an alternative dose level in the fasted state.

The optional period 4 will follow the same design as Period 3 and follow through with the follow-up phone call.



Figure 1 Study Sequence

#### 5.2 Criteria for In-Study Decisions

In-study decisions will be made by the safety advisory committee (SAC), which will always comprise the Investigator, the Sponsor's representative medical monitor or the Sponsor's medically qualified designee who is familiar with the study protocol and Investigator's Brochure (IB), and a PK expert where appropriate.

#### 5.2.1 Decision Points

The following in-study decisions will be made during this study:

- Dose level and prandial status selection for Regimen C.
- Whether to proceed with optional Period 4.
  - If Yes for Period 4, Dose level and prandial status selection for Regimen D

#### 5.2.2 Criteria for Dose Level and Prandial Status Selection

Dose level and prandial status selection for Regimen C and Regimen D (if applicable) will only be made after a complete review of all data collected from the previous dose period(s). For dose level and prandial status selection to occur, data must be available from a minimum of 12 subjects who have completed the planned PK and safety assessments up to 48 hours after dosing. If data are not available for 12 subjects, the Investigator, Scientific Lead, and Sponsor will take a decision as to whether the data available are sufficient to support the dose level and prandial status selection decision. If data in fewer subjects are used in the decision process, additional subjects will not be dosed to increase the number of subjects in the completed regimen; however, additional subjects may be enrolled to achieve the target number of subjects for subsequent regimens.

<sup>&</sup>lt;sup>a</sup> Subjects will be admitted to the clinical unit in the morning on the day before dosing (Day -1) in Period 1, and in the evening on the day before dosing (Day -1) in Period 3 and optional Period 4. Subjects will remain resident in the clinical unit between Periods 1 and 2; therefore, no admission procedures will be conducted for Period 2

b Period 4 is optional

<sup>&</sup>lt;sup>c</sup> Periods 2 to 4 only. Subjects will remain resident in the clinical unit between Periods 1 and 2; there will be a minimum washout of 4 days between dosing in Periods 1 and 2

<sup>&</sup>lt;sup>d</sup> A follow-up phone call will take place on Day 6 ± 1 of the final treatment period, to ensure the ongoing wellbeing of the subjects. If a subject reports any AEs that present a cause for concern, they will be required to attend the clinical unit for an (unscheduled) follow-up visit

Regimens C and D will only be administered in the fed state if the selected dose level has previously been administered in the fasted state.

The following data are required:

- AEs.
- Vital signs.
- ECGs.
- Safety laboratory tests.
- Plasma concentrations of delafloxacin.
- PK parameter estimates (Cmax, Tmax, AUC(0-last), AUC(0-inf) and Frel comparisons) up to 48 hours post-dose.

The dose(s) selected for Regimen C or Regimen D (if applicable) will only be selected from the design space of 300 mg to 600 mg.

The decisions on dose level and prandial status will be made by the SAC. The decision will be documented and signed by the Investigator as per Quotient Sciences' current standard operating procedure (SOP). Evidence of the decision will be retained in the ISF.

#### 5.3 Study Sample Size

The study is exploratory, and no formal sample size calculation has been made. Based on experience from previous studies of a similar design, a sample size of 16 subjects and a minimum of 12 evaluable subjects is considered sufficient to meet the objectives of the study.

#### 5.4 Randomisation (including Replacement Subjects)

Periods 1 and 2 are randomised; therefore, a randomisation schedule will be produced for these periods.

Instructions to dispense and dose will be produced prior to dosing using the randomisation schedule and will be retained in the ISF.

The original randomisation schedule and proof of quality control (QC) procedures will be held by the Data Sciences department at Quotient Sciences until the study is archived, at which time the randomisation materials will be retained in the ISF.

Using a computer-generated randomisation schedule, subject numbers will be allocated to one of two sequences in a 1:1 ratio (AB or BA [see Table 1 for regimen details]). The allocation will be balanced, with 8 subjects receiving each sequence.

Subjects will be randomised immediately prior to dosing in Period 1.

Period 3 and optional Period 4 are non-randomised; therefore, a randomisation schedule will not be produced for these periods. Instructions to dispense and dose will be produced prior to dosing with IMP, which will dictate the order in which the treatments should be administered to each subject. The instructions to dispense and dose will be retained in the ISF.

#### 5.5 Blinding Issues

This is an open-label study and therefore blinding is not required.

## 6 Populations and Analysis Sets

All safety and PK data will be presented by actual regimen received, regardless of mis-randomisation. For the statistical model, analysis set, disposition and demography tables, and listings, regimen sequence refers to the planned regimen sequence.

#### 6.1 Safety Population and Safety Analysis Set

The safety population will include all subjects who have received any amount of IMP.

The safety analysis set will be defined on a per-regimen basis and will include all safety data from the subjects included in the safety population who have received that regimen.

The safety population will be confirmed by Quotient with approval from Melinta after database lock and will be summarised for the populations table and to determine the subjects to be included in the safety analysis set.

The safety analysis set will be confirmed by Quotient with approval from Melinta at the same time as the safety population and will be summarised for the analysis of demographic and baseline characteristics, and all safety data.

#### 6.2 Pharmacokinetic Population and Pharmacokinetic Analysis Set(s)

The PK population will include all subjects who have received at least 1 dose of IMP and who satisfy the following criteria for at least 1 profile:

- No missing samples or invalid post-dose analytical results at critical time points, e.g., around Cmax
- No relevant protocol deviations that may impact the study objectives with respect to the PK endpoints
- No relevant AEs such as vomiting that suggest that the whole dose was not available for absorption for a particular subject

The PK analysis set will be defined on a per-regimen basis and will include all relevant data from the subjects included in the PK population who have received that regimen.

Individual subject profiles (i.e., regimens) will be excluded from the PK analysis set where deemed appropriate such as if the subject's data for the regimen affected did not meet the bullet point criteria above, or other study emergent point related to PK analysis or interpretation.

If required, a PK analysis subset(s) will also be documented by Quotient, with approval from Melinta, at the same time as the PK population and analysis set, if additional subjects are required to be excluded from the statistical analysis (for example to exclude subjects who have not received both the test and reference products).

The PK population will be used for the populations table. The PK analysis set and/or the PK analysis subset(s), if defined, will be used for the provision of PK summary tables and figures as well as the formal statistical analysis.

#### 6.3 Taste/Palatability Population and Taste/Palatability Analysis Set(s)

The taste population will include all subjects who have completed at least one taste test, completed at least one question on the taste questionnaire, and do not have any relevant protocol deviations.

The taste analysis set will be defined on a per-regimen basis and will include all relevant data from participants included in the taste population who have received that regimen.

The taste population will be confirmed by Quotient with approval from Melinta after database lock and will be summarised for the populations table and to determine the subjects to be included in the taste analysis set.

The taste analysis set will be confirmed by Quotient with approval from Melinta at the same time as the taste population and will be summarised for the analysis of all taste data.

# 7 Subject Disposition, Demographics and Baseline Characteristics

No formal statistical testing will be performed on subject disposition or on demographic or baseline data. Summaries of subject disposition and analyses populations will be based on all enrolled subjects. Summaries of all other data described in this section will be based on the safety analysis set unless otherwise stated. All listings will be presented by all enrolled subjects.

#### 7.1 Screening Failures

Data for subjects who have failed screening will be databased but will not be cleaned and therefore will not be included in the SDTM or ADaM datasets or any of the TFLs or the CSR.

#### 7.2 Subject Disposition and Withdrawals

The number and percentage of subjects enrolled, dosed, completed, and discontinued will be presented by sequence and overall. If any subjects discontinued from the study early then the number of subjects for each reason for discontinuation will be presented by sequence and overall. However, if none of the subjects discontinued from the study early, then the reasons for discontinuation will not be populated in the summary table. A subject may be discontinued from the study early for 1 reason only.

Subject disposition and withdrawal data will be listed, including details of informed consent.

Protocol deviations and any violations of the inclusion/exclusion criteria will also be listed.

#### 7.3 Analysis Populations

A summary table will be produced detailing the number and percentage of subjects in each population (i.e., safety, PK, and taste/palatability) by sequence and overall. The reasons for exclusion from each population will also be included in the summary table. However, if none of the subjects were excluded from a population, then the reasons for exclusion will not be populated in the summary table. A subject may be excluded from a population for more than 1 reason. The denominator for the percentage is the number of subjects enrolled in the respective sequence or overall.

Details of subjects included and excluded in the different analysis populations will be listed.

#### 7.4 Analysis Sets and Subsets

A summary table will be produced detailing the number and percentage of subjects in each of the safety, PK and taste/palatability analysis sets and analysis subset/s (if applicable) for each regimen. Separate tables will be presented for safety, PK, and taste/palatability analysis sets and each table will be based on the relevant population the analysis set is derived from. If analysis subsets are defined, they will be included on the same table as the corresponding analysis set. The reasons for exclusion from each analysis set/subset will also be included in the summary. However, if none of the subjects were excluded from an analysis set/subset, then the reasons for exclusion will not be populated in the summary table. A subject may be excluded from an analysis set/subset for more than 1 reason. The denominator for the percentage is the number of subjects in each population.

Details of subjects included and excluded in the different analysis sets/subsets will be listed.

#### 7.5 Demographic Characteristics and Lifestyle Details

Demographic data (year of birth, age, ethnicity, race, sex, height [cm], weight [kg], and body mass index [BMI; kg/m²]) will be recorded at screening.

Summary statistics (number of subjects with an observation [n], mean, standard deviation [SD], median, minimum, and maximum) will be presented for age, height, weight, and BMI at screening, by sequence and overall. The number and percentage of subjects will be presented by sequence and overall for ethnicity, race, and sex. The denominator for the percentage is all subjects in the safety analysis set for respective sequence or overall. If any values are missing, a "missing" row will be presented on the table.

Lifestyle details (i.e., smoking history [does the subject smoke, use e-cigarettes or use nicotine replacement products?] and alcohol consumption) will be summarised by sequence and overall, as categorical variables.

Demographic and lifestyle data will be listed (including weight at admission).

#### 7.6 Medical/Surgical History

Medical/surgical history will be recorded for each subject at the screening visit and updated at admission. Medical histories will be coded using MedDRA v27.0 (or a more recent version), including Lower Level Term, Preferred Term (PT), High Level Term, High Level Group Term and System Organ Class (SOC). All medical/surgical history data will be listed including coded terms (SOC and PT).

#### 7.7 Prior and Concomitant Medication

Medications (product name) will be coded using the World Health Organization (WHO) Drug Dictionary Global Drug Reference: 2024 Mar version (or more recent version), using the following Anatomical Therapeutic Chemical (ATC) classification codes:

- Product name
- Preferred name
- Drug code
- Anatomical Main Group (ATC 1<sup>st</sup> level code)
- Therapeutic subgroup (ATC 2nd level code)

- Pharmacological Subgroup (ATC 3rd level name and code)
- Chemical subgroup (ATC 4th level code)

Prior medications are defined as medications that start and stop prior to the first dose of IMP. All other medications will be defined as concomitant medications, including those that start prior to the first dose of IMP and continue thereafter. Any medications with an unknown start or stop date will be assumed to be concomitant medications, unless a partial start or stop date indicates otherwise.

All medications, including coded terms (product name, preferred term ATC 2nd level and ATC 4th level code), will be listed. One combined data listing of prior and concomitant medications will be provided. All prior medications as defined above will be flagged with a "#" symbol. Within this flagged group, medications that started after screening and stopped before dosing of IMP will also be flagged using a "\*" symbol.

#### 7.8 Other Baseline Characteristics

All other baseline characteristics, as listed below, at screening and on admission (unless otherwise stated) for each period (as appropriate) will be listed:

- Urine drug screen
- Alcohol breath test
- · Carbon monoxide test
- Virology (screening only)
- Serum pregnancy test for female subjects (screening only)
- Urine pregnancy test for female subjects (admission only)
- Follicle stimulating hormone for post-menopausal female subjects (screening only)

## 8 Efficacy

Not applicable.

#### 9 Pharmacokinetics

#### 9.1 Plasma PK Parameter Estimation

The PK parameters for delafloxacin in plasma will be estimated where possible and appropriate for each subject profile (i.e., regimen) by non-compartmental analysis methods using Phoenix WinNonlin software (v8.3 or a more recent version, Certara USA, Inc., USA). Additional parameters may be calculated if required, depending on the data.

#### 9.1.1 Definition of Plasma PK Parameters

Plasma PK parameter definitions are provided in Table 2.

Table 2 Plasma PK Parameter Definitions and Rounding Specifications

| Parameter | Definition | Unit | DP or<br>SF | No. of<br>DP/SF |
|---|---|---|---|---|
| Tlag | Time prior to the first measurable concentration | h | DP | 2 |
| Tmax | Time of maximum observed concentration | h | DP | 2 |
| Cmax | Maximum observed concentration | mass unit/mL | SF | 3 |

| Parameter | Definition | Unit | DP or<br>SF | No. of<br>DP/SF |
|---|---|---|---|---|
| AUC(0-24) | Area under the curve from time 0 to 24 h post dose | mass unit.h/mL | SF | 3 |
| AUC(0-last) | Area under the curve from time 0 to the time of last measurable concentration | mass unit.h/mL | SF | 3 |
| AUC(0-inf) | Area under the curve from time 0 extrapolated to infinity | mass unit.h/mL | SF | 3 |
| AUCextrap | Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity | % | DP | 2 |
| T1/2 | Terminal elimination half-life | h | DP | 2 |
| Lambda-z | First order rate constant associated with the terminal (log-linear) portion of the curve | 1/h | DP | 4 |
| CL/F | Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown. | mL/min | SF | 3 |
| Vz/F | Apparent volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown | L | SF | 3 |
| MRT(0-last) | Mean residence time from time 0 to time of the last measurable concentration | h | DP | 2 |
| MRT(0-inf) | Mean residence time extrapolated to infinity | h | DP | 2 |
| Frel Cmax | Relative bioavailability based on Cmax | % | DP | 2 |
| Frel AUC(0-<br>last) | Relative bioavailability based on AUC(0-last) | % | DP | 2 |
| Frel AUC(0-inf) | Relative bioavailability based on AUC(0-inf) | % | DP | 2 |
| lambda-z<br>lower* | Lower limit on time for values to be included in the calculation of lambda-z | h | DP | 2 |
| lambda-z<br>upper* | Upper limit on time for values to be included in the calculation of lambda-z | h | DP | 2 |

DP = decimal places; NA = not applicable; SF = significant figures

If 2 dose levels are administered of the same formulation in the same prandial state, then dose-normalised PK parameters will be calculated for the assessment of dose proportionality.

Dose will be used in the calculation of relevant PK parameters as per Table 3.

 Table 3
 Dose Specifications

| Dose (nominal/actual) | Nominal |
|-----------------------|-----------------|
| Precision | As per protocol |

<sup>\* =</sup> these values should be listed but omitted from the descriptive statistics

Non-dose corrected relative bioavailability (Frel) will be calculated as follows:

Frel = 
$$\left\{ \frac{\text{AUC or Cmax (test)}}{\text{AUC or Cmax (reference)}} \right\} \times 100$$

Frel will be calculated using Cmax, AUC(0-last) and AUC(0-inf). If for any reason the AUC(0-inf) is not calculable then an alternative or additional AUC over a partial area may be used to calculate Frel for all subjects.

The following comparisons will be made:

- 450 mg delafloxacin Powder for Oral Suspension (test) vs delafloxacin Tablet (reference) (Regimen A)
- 450 mg delafloxacin Powder for Oral Suspension fed (test) vs delafloxacin Powder for Oral Suspension fasted (reference)

#### 9.1.2 Rules for Plasma PK Parameter Estimation using WinNonlin

The imputation of non-numerical (e.g., below the limit of quantification [BLQ]) or negative values (e.g., pre-dose sampling times) reported in the input data set will be performed as follows for calculation of PK parameters:

- Pre-dose sample times will be entered as zero
- Values that are BLQ obtained prior to Cmax will be entered as zero
- Values that are BLQ after Cmax will be treated as missing but where BLQ concentrations are defined as parameters these will be reported as BLQ
- Values that are BLQ after Cmax may be imputed as zero for the calculation of partial AUCs, in cases where lambda-z cannot be determined
- Values that are measurable after at least 2 consecutive BLQ values after Cmax will be treated as missing for the calculation of PK parameters
- Values that are reported as "No Result" or "Not Reportable" (NR), "Not Calculated" (NC) or "No Sample" (NS) etc. will be generally be considered missing

Missing or unusual concentration values in the input data may be queried to ascertain any underlying cause. Exclusion of missing or unusual concentration values, or repeat bioanalysis of samples, will only be performed if a definitive root cause can be established and approval from Melinta Therapeutics has been obtained. Any exclusions of concentration values or repeat analysis of samples will be documented appropriately.

Plasma PK parameters will be estimated using standard Phoenix WinNonlin methods, details of which may be found in the documentation accompanying the WinNonlin software package. The rules specified in Table 4 will be applied:

Table 4 PK Parameter Estimation Details

| Sampling times | Actual |
|---|---|
| Calculation method | Linear trapezoidal linear interpolation |
| Number of points used for lambda-z | At least 3, not including Cmax |
| Minimum requirements for AUC | At least 3 consecutive measurable concentrations |

Where possible, the terminal elimination rate constant (lambda-z) will be calculated for all subject profiles. The value of lambda-z will be determined by the slope of the

regression line of the natural log transformed concentrations vs time.

The WinNonlin-determined choice of data points for determination of lambda-z will be reviewed by the pharmacokineticist, who may adjust the selection in order to provide a more appropriate fit. The choice of data points for determination of lambda-z for each profile will be confirmed following a documented peer review.

#### 9.1.3 Plasma PK Parameter Reporting Specifications

The following parameters will be reported for each regimen, as applicable, according to the rounding specifications provided in Table 1 and 2:

#### delafloxacin Tablet (reference)

g

Tlag, Tmax, Cmax, AUC(0-24), AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL/F, Vz/F, MRT(0-last), MRT(0-inf), lambda-z lower, lambda-z upper

#### delafloxacin Powder for Oral Suspension (test)

Tlag, Tmax, Cmax, AUC(0-24), AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL/F, Vz/F, MRT(0-last), MRT(0-inf), Frel Cmax<sup>a</sup>, Frel AUC(0-last)<sup>a</sup>, Frel AUC(0-inf)<sup>a</sup>, lambda-z lower, lambda-z upper

<sup>a</sup> Additional Frels based on Cmax, AUC(0-last), and AUC(0-inf) will be included, where possible, for the assessment of food effect.

The flags/footnotes given in Table 5 will be applied to the PK parameters, where relevant, and will be shown in the PK parameter listings. Additional flags may be applied based on emerging data.

| Flag | Footnote |
|---|---|
| а | Adjusted R2 of regression (the goodness of fit statistic for the elimination phase) was <0.9 |
| b | Period used for regression analysis was less than 2-fold the calculated half-life |
| С | Extrapolated portion of AUC(0-inf) >20% |
| d | Insufficient post-Cmax data points for estimation of lambda-z |
| е | Entire profile BLQ, no PK parameters could be calculated |

Table 5 PK Parameter Flags and Footnotes

In the event that the adjusted R<sup>2</sup> of regression is <0.9 ("a" flag) then lambda-z and parameter estimates derived using lambda-z and AUC(0-inf) will be deemed unreliable and will be flagged and listed but excluded from the summary statistics and formal statistical analysis.

Fewer than 3 consecutive measurable concentrations, AUCs not calculated Measurable pre-dose values were observed, however were considered less than 5 % of

Cmax

In the event that the time period used for regression analysis is less than 2-fold the calculated half-life ("b" flag) will be flagged, listed, and included in summary statistics and formal statistical analysis.

In the event that the extrapolated portion of AUC(0-inf) >20% ("c" flag), then AUC(0-inf) and parameter estimates derived using AUC(0-inf) will be deemed unreliable and will be flagged and listed but excluded from the summary statistics and formal statistical analysis.

In the event that there are insufficient post-Cmax data points for estimation of lambda-z ("d" flag) then lambda-z and parameter estimates derived using lambda-z and AUC(0-inf) will be reported as NC.

In the event that there are fewer than 3 consecutive measurable concentrations ("f" flag) then all AUC parameter estimates will be reported as NC.

In the event that measurable pre-dose values less than 5% of Cmax were observed ("g" flag), all parameter estimates for the profiles affected will be listed, flagged, and included in summary statistics and formal statistical analysis.

Note: in the event that measurable pre-dose concentrations greater than 5% of Cmax are observed, requirements for additional flags and further action will be agreed with Melinta Therapeutics and documented at the same time as the PK population.

#### 9.2 Concentration and PK Summary Tables

Summary statistics (i.e., n, mean, SD, CV%, median, minimum, maximum, geometric mean, geometric SD, and geometric CV%) of concentration data will be calculated for each time point and regimen for delafloxacin in plasma. The number of BLQ values (n#) per time point will also be presented. Geometric statistics will not be calculated for Day 1, pre-dose concentrations.

Summary statistics (i.e., n, mean, SD, CV%, median, minimum, and maximum) of plasma PK parameters will be calculated for delafloxacin for each regimen. Geometric mean, geometric SD, and geometric CV% will be presented for all plasma PK parameters except Tlag and Tmax.

Non-measurable values reported in the plasma concentration data (i.e., values that are BLQ), will be entered as zero for the determination of summary statistics, with the exception of geometric means, geometric SD, and geometric CV%, where BLQ values will be imputed as half the lower limit of quantification (LLOQ) value. Data recorded as NR, NS, or NC will be handled as missing (i.e., no assumption will be made about the actual concentration).

#### 9.3 Concentration and PK Figures

Mean, spaghetti, and individual plasma concentration vs time plots will be produced on both the linear/linear scale and log<sub>10</sub>/linear scale.

Mean plasma concentration vs time plots (using nominal times) will be produced for:

- All regimens given in the fasted state on the same plot (1 plot in total with up to 4 profiles per plot)
- Powder for Oral Suspension in the fed and fasted state for the food effect assessment on the same (1 plot in total with 2 profiles per plot).

These will be produced as follows:

- Linear/linear scale using arithmetic mean concentrations (error bars ± arithmetic SD)
- Log<sub>10</sub>/linear scale using geometric mean concentrations (error bars x/÷ geometric SD)

Separate plasma concentration vs time spaghetti plots (using actual sampling time after dosing) will be produced for each regimen with each plot displaying 1 line per subject.

Individual plasma concentration vs time plots (using actual sampling times after dosing) will be produced separately for each individual subject with all regimens on the same plot.

For all plots on a linear/linear scale, pre-dose concentration values reported as BLQ will be set to zero. Post-dose concentration values reported as BLQ will be set to zero, up to the point at which all concentrations fall below the LLOQ, after which they will be presented as missing. For all plots on a log<sub>10</sub>/linear scale, pre-dose concentration values reported as BLQ will be presented as missing. Post-dose concentration values reported as BLQ will be set to half the BLQ value, up to the point at which all concentrations fall below the LLOQ, after which they will be presented as missing. Where curves from multiple regimens or subjects are overlaid on the same plot, symbols will be used to identify different subjects/regimens and a legend will be included on the plots to define the symbols used.

#### 9.4 Concentration and PK Listings

The sample collection data (e.g., collection times) for PK samples will be listed. In addition, all concentration data and PK parameters will be listed on a per subject basis. Any flags used will be included as a footnote with the appropriate definition. Both listings will be presented by all enrolled subjects.

#### 9.5 Statistical Analysis of PK Parameters

For each analysis, distributional assumptions underlying the statistical analyses will be assessed by visual inspection of residual plots. Normality will be examined by normal probability plots, while homogeneity of variance will be assessed by plotting the residuals against the predicted values for the model. If the distributional assumptions for the parametric approach are not satisfied, then additional sensitivity analyses may be performed including the removal of potential outliers or the use of non-parametric methods to assess the robustness of the original analysis. This will be documented in the CSR together with the reasoning supporting the most appropriate action taken, if applicable. In general terms, the results of the original analysis will always be presented in the CSR.

#### 9.5.1 Relative Bioavailability

Statistical analyses will be performed on the PK parameters Cmax, AUC(0-last), and AUC(0-inf). The parameters will undergo a natural logarithmic transformation and will be analysed using a mixed effects model. The model will include terms for regimen, period and sequence as fixed effects, and subject within sequence as a random effect.

The following comparison is of interest (test vs reference):

 Regimen B (delafloxacin Powder for Oral Suspension) vs Regimen A (delafloxacin Tablet [reference])

Subjects will be included in the analysis if they have data for both test and reference in regimens included in the comparison above.

The adjusted means, including differences from the pairwise comparisons and their associated 90% CIs obtained from the model, will be back transformed on the log scale to obtain adjusted geometric mean ratios (GMRs) and 90% CIs of the ratios.

The statistical analysis will be performed using actual regimen received and planned sequence, as detailed on the randomisation schedule. The model will be fitted using the SAS Software procedure PROC MIXED. The method will be specified as Restricted Maximum Likelihood and the denominator degrees of freedom for the fixed effects will be calculated using Kenward and Roger's method [4]. The following is an example of the SAS Software code that will be used:

```
PROC MIXED DATA=<input dataset name> METHOD=REML ORDER=INTERNAL;
    CLASS TRTAN APERIODN TRTSEQPN;
    MODEL LVAR = TRTAN APERIODN TRTSEQPN / OUTP=PRED DDFM=KR;
    RANDOM SUBJIDN(TRTSEQPN);
    ESTIMATE <relevant pairwise treatment comparisons> / CL ALPHA=0.10;
    LSMEANS TRTAN / ALPHA=0.10;
    ODS OUTPUT LSMEANS=MEANS ESTIMATES=EST;
RUN;
```

#### where

- LVAR is the natural log transformed PK parameter of interest
- SUBJIDN is the numeric subject identifier variable
- TRTAN is the numeric treatment variable for the actual treatment received
- TRTSEQPN is the numeric sequence variable for the planned sequence received
- APERIODN is the numeric period variable

If there are any deviations from the planned treatment, then the analysis model specified or methods of analysis may be re-evaluated, as appropriate. Details of any deviations from the planned analysis will be documented in the CSR.

#### 9.5.2 Food Effect and Optional Dose Proportionality

Formal statistical analysis will be performed on the PK parameters Cmax, AUC(0-last), and AUC(0-inf) to assess the presence of food effect.

Additionally, formal statistical analysis will be performed on the dose-corrected PK parameters Cmax, AUC(0-last), and AUC(0-inf) to assess dose proportionality, if two dose levels of delafloxacin Powder for Oral Suspension are administered in the same prandial state.

For both food effect and dose proportionality analysis, the PK parameters will undergo a natural logarithmic transformation and will be analysed using a mixed effects model. The model will include terms for regimen as fixed effect and subject as a random effect.

The following comparisons are of interest:

- Regimen <C or D> (delafloxacin Powder for Oral Suspension Fed) vs Regimen B (delafloxacin Powder for Oral Suspension Fasted) (assessment of food effect)
- Regimen <C or D> (delafloxacin Powder for Oral Suspension yy mg) vs Regimen X (delafloxacin Powder for Oral Suspension xx mg) (where yy mg > xx mg) (optional assessment of dose proportionality)

For the assessment of food effect, subjects will be included in the analysis if they have data for both the fed and fasted state in regimens included in the comparison above.

The adjusted means, including differences from the comparisons and their associated 90% CIs obtained from the model, will be back transformed on the log scale to obtain adjusted GMRs and 90% CIs of the ratios.

The analysis will be performed using the SAS procedure PROC MIXED. The method will specified as Restricted Maximum Likelihood and the denominator degrees of freedom for the fixed effects will be calculated using Kenward-Roger method [4]. The following is an example of the SAS Software code that will be used:

- where LVAR is the natural log transformed PK parameter of interest
- SUBJIDN is the numeric subject identifier variable
- TRTAN is the numeric treatment variable for the actual treatment (i.e., prandial state or Dose) received

#### 9.5.3 Statistical Figures for Analysis of Pharmacokinetic Data

A plot of geometric mean ratios (90% CI) obtained from the statistical model to evaluate relative bioavailability and food effect will be produced for each of the PK parameters: Cmax, AUC(0-last), and AUC(0-inf), with bars representing the 90% CIs. A scatter plot will be overlayed onto the graph to show the individual ratio values.

#### 9.6 Interim PK Analysis

The details of the planned interim PK analysis are described in this section. However, as the analysis will be performed in real time, it may be necessary to change the planned analysis in response to the emerging data.

Summary tables and figures for the interim PK analysis will be presented in an Interim PK Summary Report after being exported from WinNonlin. The formatting of this output will differ slightly from the final PK output, which will be produced using SAS to include in the CSR.

The interim PK analysis will be performed on QC-checked delafloxacin concentration data in plasma using nominal sampling times and doses.

The following PK parameters will be calculated for the interim analysis:

```
<u>delafloxacin Tablet (reference)</u>
Tlag, Tmax, Cmax, AUC(0-24), AUC(0-last), AUC(0-inf), T1/2
```

#### delafloxacin Powder for Oral Suspension (test)

Tlag, Tmax, Cmax, AUC(0-24), AUC(0-last), AUC(0-inf), T1/2, Frel Cmax, Frel AUC(0-last), Frel AUC(0-inf)

#### 10 Taste Assessments

Taste will be assessed for each of the delafloxacin Powder for Oral Suspension (i.e., test) regimens administered using a questionnaire (example provided in Appendix 2) immediately following test IMP administration.

Questions 1 and 2 within the questionnaire will ask subjects to rate the acceptability of 7 taste attributes (smell, sweetness, bitterness, flavour, mouth feel/texture, and aftertaste), as well as overall acceptability on a 9-point scale. For the purposes of continuous data summaries categories on the taste scale will be assigned numerical equivalents from 1-9 where 1 = 'Dislike extremely' to 9 = 'Like extremely'. No assumption will be made for summary statistics considered missing (i.e. recorded as "not detectable") but they will be included as a category.

#### 10.1 Summary Tables for Taste Assessments

Taste assessment data for questions 1 and 2 will be summarized using descriptive statistics (i.e. n, mean, SD, minimum, Q1, median, Q3, and maximum), for overall acceptability and each taste aspect by regimen.

For each of the questions, a breakdown of the number and percentages of subjects within each rating category will also be presented by regimen (within the same table as continuous summary statistics if appropriate).

#### 10.2 Listings for Taste Assessment

All taste assessment data collected (i.e. categories for each question) will be listed for all enrolled subjects.

## 11 Safety Assessments

Safety data summaries will be presented by actual regimen and the safety analysis will be used throughout. All listing will be presented by all enrolled subjects.

#### 11.1 Extent of Exposure and Treatment Compliance

The number and percentage of subjects dosed with IMP for each regimen will be summarised.

Dosing details (including the date and time of all IMP administrations and any comments) will be listed. Any recorded deviations from the planned dosing regimen will be listed as protocol deviations.

#### 11.2 Meal Details

Meal details for fed dosing periods as recorded on the electronic case report form (eCRF) study build specification will be listed. Any recorded deviations from the planned meal times will be listed as protocol deviations.

#### 11.3 Adverse Events

Throughout the study, all adverse events (AE) will be evaluated by the PI and noted in the AE section of the eCRF study build specification. An AE is any untoward medical occurrence in a subject that occurs either before dosing (referred to as a pre-dose AE) or once a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product.

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA v27.0), and reported by system organ class (SOC) and preferred term (PT) PT.

AEs will be classified into the following categories:

- Pre-dose AEs: AEs recorded at screening or with a start date and time prior to the first dose of IMP
- Treatment-emergent adverse events (TEAEs): AEs that commence during/after the
  first dose of IMP or commence before first dose of IMP (i.e. a pre-dose AE or existing
  medical condition) but worsen in intensity during exposure to IMP

TEAEs will be assigned to the regimen of the period in which the AE first occurred. Where the severity of an AE intensifies or symptoms change in a subsequent period, this will be defined as a new AE and included under the regimen associated with the subsequent period. AEs that occur during the washout period will be assigned to the regimen the subject received during the period immediately before the washout period.

Adverse events will be classified as "mild," "moderate," or "severe" when considering their severity.

Adverse events will be classified as "unrelated", "possibly related," and "related" when considering their relationship to IMP. TEAEs classified as "possibly related" and "related" will be defined as IMP-related events. An adverse drug reaction (ADR) is any AE where a causal relationship with the IMP is at least reasonable possibility, i.e., "possibly related" and "related". Pre-dose AEs will always have the classification of "unrelated".

If the severity or relationship to IMP of a TEAE is missing, the severity/relationship will be tabulated as "missing" in the summary tables.

When summary presentation is made by maximum severity, "missing" will be handled as follows:

- If there are other events (i.e., same SOC and PT code) with a maximum severity recorded as "moderate" or "severe" for that subject and regimen, then the maximum observed severity for that subject will be categorised and presented as "moderate" or "severe", respectively
- If there are other events (i.e., same SOC and PT code) with a maximum severity recorded as "mild" for that subject and regimen, then the maximum observed severity for that subject will be categorised and presented as "missing"

When summaries are presented by relationship to regimen, "missing" will be handled as follows:

- If there are other events (i.e., same SOC and PT code) with a most closely related association recorded as "possibly related" or "related" for that subject and regimen, then the maximum observed relationship for that subject will be categorised and presented as "possibly related" or "related", respectively.
- If there are other events (i.e., same SOC and PT code) with a most closely related association recorded as "unrelated" for that subject and regimen, then the maximum observed relationship for that subject will be categorised and presented as "missing".

Where the start date of an AE is missing and the stop date is on or after the day of first administration of test-product, or both the start and stop dates are missing, then a "worst-case" scenario will be assumed i.e., the AE is assumed to have occurred post-administration and is therefore considered treatment-emergent. If a partial start date/time is available, then the event will be considered as treatment-emergent, unless the partial information suggests otherwise.

#### 11.3.1 Summary Tables for Adverse Events

All pre-dose AEs (as defined in Section 11.3) will be excluded from the summary tables, but will be listed.

Descriptive statistical methods will be used to summarise the TEAE data.

The number and percentage of subjects reporting each TEAE will be presented for both SOC and PT. For summaries by SOC and PT, with the exception of TEAEs by severity and relationship to IMP, the number of subjects, and the number of events will be summarised. For summaries by severity and relationship, only the number of subjects will be summarised.

For counts of subjects experiencing events the following will apply:

- A subject experiencing TEAEs in more than one body system, within a study period, will be counted once in the total number of subjects with TEAEs in that study period
- A subject with more than 1 TEAE in the same SOC, within a study period, counts only once at the SOC level
- A subject with more than 1 TEAE in the same PT, within a study period, counts only once at the PT level

For TEAE event counts, all events are included.

When it is necessary to calculate percentages, the denominator will be the total number of subjects in the safety analysis set for that regimen or study period and the numerator will be the total number of subjects reporting a TEAE within the relevant category.

Summaries presented for SOC and PT will be presented in descending order of frequency overall i.e. most frequently reported SOC in the study and then by most frequently reported PT in the study within each SOC.

#### 11.3.1.1 Overall Summary of Adverse Events

The following will be summarised by regimen and overall for the safety analysis set:

- Number and percentage of subjects reporting TEAEs
- Number and percentage of subjects reporting severe TEAEs
- Number and percentage of subjects reporting ADRs
- Number and percentage of subjects reporting serious TEAEs
- Number and percentage of subjects reporting TEAEs leading to subject withdrawal
- Number and percentage of subjects reporting TEAEs leading to death
- Total number of TEAEs
- Total number of severe TEAEs
- Total number of IMP-related ADRs

- Total number of serious TEAEs
- Total number of TEAEs leading to subject withdrawal
- Total number of TEAEs leading to death

### 11.3.1.2 Summary of Treatment-Emergent Adverse Events

All subjects reporting TEAEs will be summarised by regimen and overall. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 TEAE within a regimen/overall will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by regimen and overall. Counts will be given for number of subjects and number of events.

#### 11.3.1.3 Summary of Treatment-Emergent Adverse Events by Severity

All subjects reporting TEAEs will be summarised by severity (i.e. mild, moderate, or severe) and regimen. Counts will be given for number of subjects, not number of events. Counts will be given by maximum severity (i.e., subjects experiencing more than 1 TEAE within a regimen will be counted only once using the most severe episode).

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by maximum severity (i.e., mild, moderate, or severe) and regimen. Counts will be given for total number of subjects, not for events. Counts by maximum severity will be given (i.e., subjects experiencing more than 1 TEAE within a regimen will be counted only once within each SOC and PT using the most severe episode).

## 11.3.1.4 Summary of Treatment-Emergent Adverse Events by Relationship to IMP

All subjects reporting TEAEs will be summarised by relationship to IMP (i.e., unrelated, possibly related, or related) and regimen. Counts will be given for number of subjects, not number of events. Counts will be given by the closest relationship to IMP (i.e., subjects experiencing more than 1 TEAE within a regimen will be counted only once using the most closely related event).

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by closest relationship to IMP (i.e. unrelated, possibly related, or related) and regimen. Counts will be given for total number of subjects, not for events. Counts by closest relationship will be given (i.e., subjects experiencing more than 1 TEAE within a regimen will be counted only once within each SOC and PT using the most closely related event).

#### 11.3.1.5 Summary of Adverse Drug Reactions (ADRs)

All subjects reporting ADRs will be summarised by regimen. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 ADR within a regimen will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting ADRs will be summarised for SOC and PT by regimen. Counts will be given for number of subjects and number of events.

#### 11.3.1.6 Summary of Serious Adverse Events

All subjects reporting treatment-emergent serious adverse events (SAEs) will be summarised by regimen. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 SAE within a regimen will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting treatment-emergent SAEs will be summarised for SOC and PT by regimen. Counts will be given for number of subjects and number of events.

#### 11.3.2 Listings for Adverse Events

All pre-dose AEs (as defined in Section 11.3) will be listed including SOC and PT.

A separate data listing of all TEAEs will be provided including the SOC and PT. In addition, a listing of all SAEs will be provided.

#### 11.4 Laboratory Evaluations

The details of sample collection for laboratory safety analysis are described in the study protocol.

Where a value is provided by the safety laboratory as either above or below the limit of detection (LOD), this will be set to the respective LOD itself for descriptive summaries. No imputations will be made in the individual listings.

#### 11.4.1 Summary Tables for Laboratory Evaluations

Haematology and clinical chemistry data will be summarised (n, mean, SD, median, minimum, and maximum) for each laboratory parameter at each time point, including changes from baseline (Day -1, Admission for Period 1 and Day 1, Pre-dose for Periods 2 to 4) at each scheduled post-baseline time point by regimen.

Shift tables from baseline to each scheduled post-baseline time point (with respect to the number and percentage of subjects with values below, within or above the reference range) will be presented by regimen. Percentages will be based on the number of subjects with measurements at baseline and the relevant post-baseline time point.

For fasting-sensitive laboratory parameters (i.e., glucose), results taken in the non-fasted state (i.e., LBFAST=N) will not be included in summary statistics by time point or be used in derivations of changes from baseline. For tabulations (e.g., shift tables), both fasted and non-fasted results will be pooled and used in the tabulations, using the appropriate fasted or non-fasted reference range. All results (fasted or non-fasted) will be listed with non-fasted data flagged.

Reference ranges for each laboratory parameter will be presented for the relevant parameter in each summary table.

#### 11.4.2 Listings for Laboratory Evaluations

The sample collection data (e.g., collection times) for laboratory analysis and urinalysis data will be listed.

All individual subject data for planned haematology, clinical chemistry, and urinalysis data, including derivations, such as change from baseline, will be listed. If applicable, data from unscheduled laboratory tests will also be listed and flagged with a "#" to indicate that it will not be used in the summary statistics. In these listings, individual data will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively.

Separate listings of all haematology, clinical chemistry, and urinalysis values outside their reference ranges by subject will also be provided. Reference ranges will be supplied by the safety laboratory for haematology and clinical chemistry and per the eCRF for urinalysis (i.e., a positive or negative result) with the exception of the following reference ranges for urinalysis:

pH: 5.0 to 9.0

Specific gravity: 1.000 to 1.030

#### 11.5 Vital Signs

The details of measurement of vital signs (i.e., systolic and diastolic BP, heart rate, oral body temperature, respiratory rate, and clinical assessment and findings) are described in the study protocol.

#### 11.5.1 Summary Tables for Vital Signs

Vital signs data, including change from baseline (Day 1, pre-dose for each study period), will be summarised (i.e. n, mean, SD, median, minimum, and maximum) at each post-baseline time point by regimen.

In addition, the number of subjects with 'substantial' increases or decreases or no substantial change from baseline in systolic BP (>20 mmHg), diastolic BP (>10 mmHg) and heart rate (>15 bpm) will be summarised.

#### 11.5.2 Listings for Vital Signs

All individual vital signs data, including derivations, such as change from baseline, will be listed. Individual data will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively, and subjects with 'substantial' increases or decreases from baseline (as defined in Section 11.5.1) in systolic BP, diastolic BP, and heart rate will be flagged with an 'I' (increase) or 'D' (decrease), respectively. If applicable, data from unscheduled vital signs assessments will also be listed and flagged with a "#" to indicate it will not be used in the summary statistics.

In addition, a separate listing of all vital signs data outside their reference ranges by subject will also be provided.

The reference ranges (from Quotient SOP "The Interpretation of the Electrocardiogram, Vital Signs and Clinical Laboratory Data During Phase I") defined in Table 6 will be used.

Table 6 Vital Signs Reference Ranges

| Parameter | Split | Lower limit | Upper limit |
|-----------------------|-------------|----------------|----------------|
| Systolic BP | 18-45 years | 90 mmHg | 140 mmHg |
| Systolic BP | >45 years | 90 mmHg | 160 mmHg |
| Diastolic BP | NA | 40 mmHg | 90 mmHg |
| Heart rate | NA | 45 bpm | 100 bpm |
| Oral Body Temperature | NA | 35.5°C | 37.5°C |
| Respiration Rate | NA | 10 breaths/min | 24 breaths/min |

NA=Not applicable

#### 11.6 ECGs

The details of measurement of supine ECG parameters (i.e., ventricular rate, RR interval, QT interval, corrected QT interval by Fridericia's formula (QTcF), PR Interval, QRS duration, QRS axis, rhythm, interpretation, and clinical significance and findings) are described in the study protocol.

#### 11.6.1 Summary Tables for ECGs

ECG data, including change from baseline (Day 1, pre-dose for each study period), will be summarised (i.e., n, mean, SD, median, minimum, and maximum) at each post-baseline time point by regimen.

The number and percentage of subjects with normal and prolonged QTcF and increases in QTcF intervals from baseline within the categories defined in Table 7 (based on the International Council on Harmonisation [ICH] E14 guideline [5]) will be summarised by time point. Percentages will be based on the number of subjects with measurements at the relevant time point.

Table 7 ICH E14 Ranges for QTcF

| Parameter | ICH E14 Range |
|--------------------------------|--------------------|
| | ≤450 msec (normal) |
| QTcF | 451-480 msec |
| | 481-500 msec |
| | >500 msec |
| | ≤30 msec |
| Increase in QTcF from baseline | 31-60 msec |
| | >60 msec |

#### 11.6.2 Listings for ECGs

All ECG measurements (i.e., single readings), including derivations, such as change from baseline, will be listed.

All ECG measurements will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively. If applicable, data from unscheduled ECG assessments will also be listed and flagged with a "#" to indicate that it will not be used in the summary statistics.

In addition, measurements with increase in QTcF from baseline of 31-60 msec and with 'substantial increases' (>60 msec) will be flagged with 'l' and 'Sl', respectively.

Separate listings of all ECG parameters outside their reference range by subject and also with QTcF increases from baseline >30 msec will also be provided.

The reference ranges (from the eCRF study build specification for all parameters, except QT Interval, which is from Quotient SOP "The Interpretation of the Electrocardiogram, Vital Signs and Clinical Laboratory Data During Phase I / II Clinical Trials") and defined in Table 8 will be used.

Table 8 ECG Reference Ranges

| Parameter | Split | Lower limit | Upper limit |
|------------------|---------|-------------|-------------|
| Ventricular Rate | NA | 45 bpm | 100 bpm |
| QT Interval | NA | NA | 500 msec |
| QTcF Interval | Males | NA | 450 msec |
| QTcF | Females | N/A | 470 msec |
| PR Interval | NA | 120 msec | 220 msec |
| QRS Duration | NA | NA | 120 msec |
| QRS Axis | NA | -30° | 100° |
| RR Interval | N/A | 600 msec | 1333 msec |

NA=Not applicable

#### 11.7 Physical Examination

All physical examination details and comments on any physical examination findings will be listed.

## 12 Interim Statistical Analyses

No interim statistical analysis is planned for this study.

## 13 Changes in the Conduct of the Study or Planned Analysis

#### 13.1 Changes in the Conduct of the Study

No changes in the conduct of the study had been reported at the time this document was written.

#### 13.2 Changes to the Planned Analyses

No changes to planned analysis.

#### 13.3 Any Other Relevant Changes

Not applicable.

#### 14 Overall Considerations

#### 14.1 Statistical Programming and Analysis

The Data Sciences Department at Quotient will perform the statistical programming and analysis to produce all analysis datasets and TFLs using the statistical SAS Software v9.4 (or more recent version).

In general terms, categorical data will be presented using counts and percentages, while continuous variables will be presented using n, mean, SD, median, minimum, and maximum. For PK data, additional statistics including CV%, geometric mean, geometric SD, and geometric CV% will be presented, as appropriate.

The geometric mean is obtained by applying a natural log transformation to the raw data, calculating the arithmetic mean of the transformed values and then back transforming the arithmetic mean.

The following formula will be used to calculate the geometric SD:

i.e., a natural log transformation is applied to the raw data, the arithmetic SD of the transformed values is calculated, and then the arithmetic SD of the transformed values is back transformed.

The following formula will be used to calculate the geometric CV%:

geometric CV% = 
$$100 \times (\exp{SD[(\log(\text{raw data})]}^2 - 1)^{1/2}$$

i.e., a natural log transformation is applied to the raw data, the arithmetic SD of the transformed values is calculated. This value is then squared. The square value is back transformed and a value of 1 is subtracted from the back transformed value. A square root is then applied and the resulting value is multiplied by 100.

In general summary statistics and statistical analysis results will be presented as detailed in Table 9, unless otherwise stated:

**Table 9 Reporting Conventions for Summary Statistics and Statistical Analysis** 

| Data Type | Statistic | Number of decimal places for reporting (i) |
|---|---|---|
| Frequency | Counts (n) | None |
| | Percentages (%) | 1 decimal place |
| | n | None |
| | Mean | i + 1 decimal places |
| | Median | i + 1 decimal places |
| | SD | i + 1 decimal places |
| | Min | i decimal places |
| Summary statistic | Max | i decimal places |
| | Q1 | i decimal places |
| | Q3 | i decimal places |
| | CV% | 1 decimal place |
| | Geometric Mean | i + 1 decimal places |
| | Geometric SD | i + 1 decimal places |
| | Geometric CV% | 1 decimal place |
| Statistical analysis | Ratios (%) | 2 decimal places |
| | Ratios * | 3 decimal places |
| | Confidence intervals (%) | 2 decimal places |
| | Confidence intervals * | 3 decimal places |
| | | if <0.001: presented as <0.001 |
| | p-values | if ≥0.001 and <0.099: presented to 3 decimal places |
| | | all other p-values will be presented to 2 decimal places |

i refers to the number of decimal places reported in the eCRF or other appropriate source data for the original data. Where bioanalytical or PK data are received rounded in significant figures rather than decimal places, summary statistics will be supplied to the same precision.

\* Where ratios are not presented as (%) (e.g., optional assessment of dose proportionality)

Details of how the individual PK parameters will be presented are detailed in Section 9.1.1. Where data requires rounding, values ending with 1 to 4 will be rounded down and values ending with 5 to 9 will be rounded up.

All data listings will be based on all enrolled subjects (as defined in Section 3.2.1). Details of age and sex will be included on all data listings.

All statistical tests relating to PK parameters will be 2-sided and will be performed using a 10% significance level, leading to 90% (2-sided) confidence intervals (CIs).

If any baseline measurements are found to be missing then consideration will be given to imputation using the preceding time point (e.g., screening, admission, if applicable). Unscheduled assessment may be used if appropriate. Details of any such imputations will be documented as part of the safety analysis set.

There will be no other imputations for the safety data with regard to missing values or study discontinuation (i.e., subjects who do not complete the study). Imputation for PK parameter estimation using WinNonlin is described in Section 9.1.2 and for reporting PK data is described in Section 9.1.3.

If partial dates are available for smoking history, prior medications, or medical/surgical history, there will be no date imputations. The data listings will only show the date information for the date part that is available (e.g., if only the year part of the date is available then YYYY will be presented in the listing). If the full date information is missing, then this will be presented as missing on the data listing.

If the start date/time of an AE record is missing or incomplete, preventing a clear allocation of the AE to a single treatment period, a worst-case consideration (see below) will be done aiming to allocate the AE record to one single treatment period, if possible. When a worst-case consideration is needed, any available start or end date/time will be considered in assignment of the AE to a treatment period.

- An AE which according to the available information of its start date/time could belong to screening as well as to the first treatment period will only be placed in the first treatment period
- An AE which according to the available information of its start date/time could belong to two (or more) subsequent treatment periods will be allocated to all the matching treatment periods (i.e., these AE records will be replicated and reported once in each of these matching treatment periods where IMP was administered before the end date)
- An AE which according to the available information of its start date/time could belong to all possible treatment periods will be allocated to all the treatment periods
# 14.2 Quality Control of Summary Tables, Figures and Listings and Statistical Analysis

Isolated data errors detected as a result of the QC checks that are deemed significant (i.e., errors that would impact the interpretation of the results in relation to the study objectives) will be corrected as per the data management plan. Systematic data errors will be investigated further. The data will be corrected if necessary, and the appropriate table, figure, and/or listing re-generated and then re-checked.

In addition to QC checks, a documented peer review will be performed of all SAS Software-generated report standard TFLs, including a review of SAS Software code and program log files.

## 14.2.1 Quality Control - Summary Tables

Manual QC methods (i.e., comparison of results in the table to results calculated by a calculator or spreadsheet) will be used for all analyses and summary tables. All summary tables will be QC'd as follows:

- Where tables are presented by regimen (i.e., no time points), QC will alternate between regimen to avoid the same regimen being QC'd every time. For tables presented by regimen only (i.e., no time points), all summary statistics for 1 regimen will be QC'd
- Where tables are presented by regimen and time point, QC will alternate between regimen and time point, to avoid the same regimen being QC'd every time
- For tables presented by regimen and time point, a single regimen at 1 time point in each table will be QC'd
- Where tables are produced using a macro for multiple parameters, a minimum of 3 tables, using different regimens or combinations of regimens and time point as appropriate, will be QC'd
- For AEs, the treatment details will be 100% QC'd against the randomisation schedule (If applicable) for all subjects
- AE summary tables will be 100% checked using the relevant data listing

### 14.2.2 Quality Control - Figures

All figures will be QC'd manually using the corresponding/appropriate summary table or data listing, as follows:

- Across all figures, QC will alternate between regimen, to avoid the same regimen being QC'd every time
- Where a figure presents data from more than 1 regimen, only 1 regimen will be QC'd.
   However, all data points for that regimen will be checked
- Where figures are produced using a macro for individual subjects and/or multiple parameters, a minimum of 3 figures will be QC'd
- Mean figures will be QC'd using the corresponding summary table
- Figures showing individual data will be QC'd using the corresponding data listing

## 14.2.3 Quality Control - Data Listings

All data listings will be subjected to a 100% manual check against the eCRF study build specifications or other appropriate source data for a minimum of 2 subjects. If appropriate, the subjects checked will include at least 1 subject who withdrew early from the study.

The study treatment allocation details on the dosing data listing will be 100% QC checked against the study randomisation schedule.

## 14.2.4 Quality Control - Statistical Analysis

QC of statistical analyses will be performed by peer review of program code, log, and output. This will be performed by a statistician at Quotient who is not responsible for performing the statistical analysis.

### 15 SAS Data Transfer

All study data used for analysis and reporting will be transferred to Melinta on issue of the final CSR. Datasets will be provided in SAS transport file format (XPT). Each dataset will be an individual transport file and will be performed in compliance with ADaM (IG v1.1). This will include define.xml (v2.0) output as well as a Data Reviewers Guide (adrg) in PDF format which will be linked to the define.xml. There will be one draft transfer ADaM define.xml and one final, issued on finalisation of the CSR.

Details of the SDTM define.xml are documented in the study Data Management Plan.

## 16 Programming Conventions

Quotient standards for layout of TFLs and programming conventions will be used as follows:

- Courier new, font size 8
- Landscape
- A4 paper
- US letter size (8.5 x 11)

Tables and listings will be produced as MS Word 2016 (or more recent version) documents and figures will be produced as PDF files. Listings will be sorted by subject ID and period (where applicable), i.e., all subjects will be presented in sequential order, and then chronologically within each subject where both periods are presented; treatment sequence will be displayed for listings where no period is required to be presented.

The mock tables (Section 21), figures (Section 22), and data listings (Section 23) presented are a representation of Quotient reporting standards. However, these are provided for illustrative purposes only. The numbering and titles, formatting, labelling, footnotes, and cosmetic appearance of all output may be modified or additional labelling/footnotes may need to be added during analysis and reporting, for clarification purposes. Any such changes will not be regarded as changes to planned analyses.

### 17 Reference List

- [1] Gough K, Hutchison M, Keene O, et al. Assessment of dose proportionality: report from the statisticians in the pharmaceutical industry/pharmacokinetics UK joint working party. *Drug Info J.* 1995; 29(3): 1039–1048
- [2] Smith BP, Vandenhende FR, DeSante KA, et al. Confidence interval criteria for assessment of dose proportionality. *Pharmaceutical Research*. 2000; 17(10): 1278–1283.

- [3] Hummel J, McKendrick S, Brindley C, et al. Exploratory assessment of dose proportionality: review of current approaches and proposal for a practical criterion. *Pharmaceutical Statist*. 2009; 8: 38–49
- [4] Brown, Prescott. Repeated measures data. In: Brown H and Prescott R, 3<sup>rd</sup> edition. *Applied Mixed Models in Medicine*. Chichester, UK: John Wiley & Sons Ltd; 2015: 242–243.
- [5] International Council for Harmonisation (ICH) Topic E 14, The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs Guidelines approved by the Committee for Medicinal Products for Human Use (CHMP) in May 2005 which came into force November

## 18 Index of Tables

| Table<br>Number | Table Title |
|---|---|
| | Subject Disposition, Populations and Datasets |
| 14.1.1 | Subject Disposition by Reason<br>Summary Statistics: All Enrolled Subjects |
| 14.1.2.1 | Analysis Populations<br>Summary Statistics: All Enrolled Subjects |
| 14.1.2.2 | Safety Analysis Set<br>Summary Statistics: All Enrolled Subjects |
| 14.1.2.3 | PK Analysis Set/Subset<br>Summary Statistics: All Enrolled Subjects |
| 14.1.2.4 | Taste/Palatability Analysis Set<br>Summary Statistics: All Enrolled Subjects |
| | Demographic and Baseline Characteristics |
| 14.1.3 | Demographic and Baseline Characteristics<br>Summary Statistics: Safety Analysis Set |
| 14.1.4 | Lifestyle Details: Smoking History and Alcohol Consumption Summary Statistics: Safety Analysis Set |
| | Dosing Details |
| 14.1.5 | Extent of Exposure<br>Summary Statistics: Safety Analysis Set |
| | Plasma Pharmacokinetic Concentrations |
| 14.2.1 | Plasma Pharmacokinetic Concentrations<(units)>: Delafloxacin Summary Statistics: PK Analysis Set |
| 14.2.2 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Summary Statistics: PK Analysis Set |
| 14.2.3.1 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Statistical Analysis Results – Assessment of Relative Bioavailability: PK<br>Analysis Set |
| 14.2.3.2 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Statistical Analysis Results – Assessment of Relative Bioavailability Fixed<br>Effects Table: PK Analysis Set |
| 14.2.3.3 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Statistical Analysis Results – Assessment of Food Effect: <pk <br="" analysis="" set="">PK Analysis Subset&gt;</pk> |
| 14.2.3.4 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Statistical Analysis Results – Assessment of Dose Proportionality PK<br>Analysis Set<br>Programming note: Optional table |
| | Taste Assessments |

| Table<br>Number | Table Title |
|---|---|
| 14.2.4 | Taste Assessments Summary Statistics: Taste/ Palatability Analysis Set <overall acceptability="" aspect="" taste=""></overall> |
| | Adverse Events |
| 14.3.1 | Overall Summary of Treatment-Emergent Adverse Events Summary Statistics: Safety Analysis Set |
| 14.3.2 | Treatment-Emergent Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set |
| 14.3.3 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Severity Summary Statistics: Safety Analysis Set |
| 14.3.4 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Relationship to IMP Summary Statistics: Safety Analysis Set |
| 14.3.5 | Adverse Drug Reactions By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set |
| 14.3.6 | Serious Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set |
| | Laboratory Results |
| 14.4.1 | Haematology Summary Statistics: Safety Analysis Set Parameter <units></units> |
| 14.4.2 | Haematology<br>Shift Analysis: Safety Analysis Set<br>Parameter <units></units> |
| 14.4.3 | Clinical Chemistry Summary Statistics: Safety Analysis Set Parameter <units></units> |
| 14.4.4 | Clinical Chemistry Shift Analysis: Safety Analysis Set Parameter <units></units> |
| | Vital Signs and ECG Results |
| 14.5.1 | Vital Signs Summary Statistics: Safety Analysis Set Parameter <units></units> |
| 14.5.2.1 | ECGs Summary Statistics: Safety Analysis Set Parameter <units></units> |

| Table<br>Number | Table Title |
|---|---|
| | ECGs QTcF Categorical Data Summary Statistics: Safety Analysis Set |

# 19 Index of Figures

| Figure<br>Number | Figure Title |
|---|---|
| | Plasma Pharmacokinetic Concentrations |
| 14.2.1.1 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Linear/Linear Scale Arithmetic Mean (±Arithmetic SD) Values: <pk analysis="" pk="" set="" subset=""> All Fasted Regimens</pk> |
| 14.2.1.2 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Log10/Linear Scale Geometric Mean (×/÷ Geometric SD) Values: <pk analysis="" pk="" set="" subset=""> All Fasted Regimens</pk> |
| 14.2.1.3 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Linear/Linear Scale Arithmetic Mean (±Arithmetic SD) Values: <pk analysis="" pk="" set="" subset=""> Fed vs Fasted Comparison</pk> |
| 14.2.1.4 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Linear/Linear Scale Arithmetic Mean (±Arithmetic SD) Values: <pk analysis="" pk="" set="" subset=""> Fed vs Fasted Comparison</pk> |
| 14.2.2.1 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Linear/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" pk="" set="" subset=""> <regimen></regimen></pk> |
| 14.2.2.2 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Log10/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" pk="" set="" subset=""> <regimen></regimen></pk> |
| 14.2.3.1 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Linear/Linear Scale Individual Values for Subject <xxx>: <pk analysis="" pk="" set="" subset=""></pk></xxx> |
| 14.2.3.2 | Plasma Pharmacokinetic Concentrations: Delafloxacin (units) Log10/Linear Scale Individual Values for Subject <xxx>: <pk analysis="" pk="" set="" subset=""></pk></xxx> |

| Figure<br>Number | Figure Title |
|---|---|
| | Statistical Plots |
| 14.2.4.1 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Log10/Log10 Scale<br>Individual and Mean (×/÷Geometric SD) Values – Relative<br>Bioavailability: PK <pk analysis="" pk="" set="" subset=""></pk> |
| 14.2.4.2 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Log10/Log10 Scale<br>Individual and Mean (×/÷Geometric SD) Values – Food Effect: PK <pk<br>Analysis Set/PK Analysis Subset&gt;</pk<br> |

# 20 Index of Listings

| | - Liotingo |
|---|---|
| Listing<br>Number | Listing Title |
| | Subject Informed Consent and Completion/Withdrawal |
| 16.2.1 | Subject Informed Consent and Completion/Withdrawal Individual Values: All Enrolled Subjects |
| | Protocol Deviations and Inclusion/Exclusion Criteria |
| 16.2.2.1 | Protocol Deviations<br>Individual Values: All Enrolled Subjects |
| 16.2.2.2 | Inclusion/Exclusion Criteria<br>Individual Values: All Enrolled Subjects |
| | Analysis Populations and Reasons for Exclusion |
| 16.2.3.1 | Analysis Populations and Reasons for Exclusion Individual Values: All Enrolled Subjects |
| 16.2.3.2 | Analysis Sets and Analysis Subsets and Reasons for Exclusion Individual Values: All Enrolled Subjects |
| | Demographic and Baseline Characteristics |
| 16.2.4.1 | Demographics and Baseline Characteristics<br>Individual Values: All Enrolled Subjects |
| 16.2.4.2 | Lifestyle Details: Smoking History and Alcohol Consumption Individual Values: All Enrolled Subjects |
| 16.2.4.3 | Medical/Surgical History<br>Individual Values: All Enrolled Subjects |
| 16.2.4.4 | Prior and Concomitant Medication<br>Individual Values: All Enrolled Subjects |
| 16.2.4.5 | Urine Drug Screen<br>Individual Values: All Enrolled Subjects |
| 16.2.4.6 | Alcohol Breath and Carbon Monoxide Test<br>Individual Values: All Enrolled Subjects |
| 16.2.4.7 | Virology<br>Individual Values: All Enrolled Subjects |
| 16.2.4.8 | Urine/Serum Pregnancy Test<br>Individual Values: All Enrolled Female Subjects |
| 16.2.4.9 | Follicle Stimulating Hormone<br>Individual Values: All Enrolled Post-Menopausal Female Subjects |
| | Dosing Details and Meal Details |
| 16.2.5.1.1 | Dosing Details<br>Individual Values: All Enrolled Subjects |
| 16.2.5.1.2 | Meal Details for Fed Dosing<br>Individual Values: All Enrolled Subjects |

| Listing<br>Number | Listing Title |
|---|---|
| | Plasma Pharmacokinetic Concentration and Parameters |
| 16.2.5.2 | Blood Sample Collection Details for Pharmacokinetic Analysis and Plasma Concentrations: Delafloxacin Individual Values: All Enrolled Subjects |
| 16.2.6.1 | Plasma Pharmacokinetic Parameters: Delafloxacin<br>Individual Values: All Enrolled Subjects |
| | Taste Assessment |
| 16.2.6.2 | Taste Assessment<br>Individual Values: All Enrolled Subjects |
| | Adverse Events |
| 16.2.7.1 | Pre-dose Adverse Events<br>Individual Values: All Enrolled Subjects |
| 16.2.7.2 | All Treatment-Emergent Adverse Events Individual Values: All Enrolled Subjects |
| 16.2.7.3 | Serious Adverse Events<br>Individual Values: All Enrolled Subjects |
| | Laboratory Data |
| 16.2.8.1 | Blood Sample Collection Details for Laboratory Analysis<br>Individual Values: All Enrolled Subjects |
| 16.2.8.2 | Haematology<br>Individual Values: All Enrolled Subjects |
| 16.2.8.3 | Haematology<br>Individual Values Outside the Reference Range: All Enrolled Subjects |
| 16.2.8.4 | Clinical Chemistry<br>Individual Values: All Enrolled Subjects |
| 16.2.8.5 | Clinical Chemistry<br>Individual Values Outside the Reference Range: All Enrolled Subjects |
| 16.2.8.6 | Urinalysis Sample Collection<br>Individual Values: All Enrolled Subjects |
| 16.2.8.7 | Urinalysis<br>Individual Values: All Enrolled Subjects |
| 16.2.8.8 | Urinalysis<br>Individual Values Outside the Reference Range: All Enrolled Subjects |
| | Vital Signs and ECGs |
| 16.2.9.1.1 | Vital Signs<br>Individual Values: All Enrolled Subjects |
| 16.2.9.1.2 | Vital Signs<br>Individual Values Outside the Reference Range: All Enrolled Subjects |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.9.2.1 | ECGs<br>Individual Values: All Enrolled Subjects |
| 16.2.9.2.2 | ECGs<br>Individual Values Outside the Reference Range: All Enrolled Subjects |
| | Other Data |
| 16.2.9.3 | Physical Examination Data<br>Individual Values: All Enrolled Subjects |

## 21 Mock Tables

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.1.1

Subject Disposition by Reason

Summary Statistics: All Enrolled Subjects

#### Sequence

| | ABC <d> (N=X) n (%)</d> | BAC <d><br/>(N=X)<br/>n (%)</d> | Overall (N=X) n (%) |
|---|---|---|---|
| Subjects enrolled (1) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects dosed | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects completed | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for discontinuation | | | |
| REASON 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| REASON 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| REASON 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> (1) An enrolled subjects signed the informed consent, qualified per the inclusion/exclusion criteria and was randomised A subject may be discontinued for one reason only

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all reasons for discontinuation as recorded on the source. If none of the subjects discontinued from the study early then reasons for discontinuation will not be populated in the summary table

Percentages are based on the number of subjects enrolled in the respective sequence

Melinta Therapeutics
Protocol: ML-DEL-101-3727-1

Page x of y

TABLE 14.1.2.1
Analysis Populations
Summary Statistics: All Enrolled Subjects

#### Sequence

| | ABC <d> (N=X) n (%)</d> | BAC <d><br/>(N=X)<br/>n (%)</d> | Overall (N=X) n (%) |
|---|---|---|---|
| Subjects in safety population Reason for exclusion from safety population | , , | xx (xx.x) | , , |
| <pre><all categories="" listing="" on="" source=""></all></pre> | xx (xx.x)<br> | xx (xx.x)<br> | xx (xx.x)<br> |
| Subjects in PK population Reason for exclusion from PK population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre><all categories="" listing="" on="" source=""></all></pre> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects in taste/palatability population Reason for exclusion from taste/palatability population | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) |
| <pre><all categories="" listing="" on="" source=""></all></pre> | xx (xx.x)<br> | xx (xx.x)<br> | xx (xx.x)<br> |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> A subject may be excluded for more than one reason

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: Percentages are based on the number of subjects enrolled in the respective sequence

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.1.2.2 Safety Analysis Set

Summary Statistics: Safety Population

| | 450 MG TAB<br>FASTED<br>(N=X)<br>n (%) | 450 MG POS<br>FASTED<br>(N=X)<br>n (%) | XXX MG POS <status> (N=X) n (%)</status> | XXX MG POS <status> (N=X) n (%)</status> |
|---|---|---|---|---|
| Subjects in safety analysis set Reasons for exclusion from safety analysis set | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre><all categories="" from="" source=""></all></pre> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> A subject may be excluded for more than one reason

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: A similar table will be produced for the PK Analysis Set and Taste/palatability Analysis Set (and Subset[s], if required), i.e. Table [14.1.2.3] and Table [14.1.2.4]

Each analysis set/subset will be a subset of their respective population and percentages

will be based on number of subjects in each population

Melinta Therapeutics
Protocol: ML-DEL-101-3727-1

Page x of y

TABLE 14.1.3

Demographic and Baseline Characteristics Summary Statistics: Safety Population

#### Sequence

| | | ABC <d> (N=X)</d> | BAC <d></d> | Overall (N=X) |
|---|---|---|---|---|
| Age (years) | n<br>Mean<br>SD<br>Median<br>Min<br>Max | XX<br>XX.XX<br>XX.XX<br>XX.X<br>XX.X | xx<br>xx.xx<br>xx.xx<br>xx.xx<br>xx.xx<br>xx.x | xx<br>xx.xx<br>xx.xx<br>xx.xx<br>xx.xx<br>xx.x |
| Ethnicity n(%) | <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race n(%) | <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sex n(%) | Male<br>Female | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | , , |
| Height (cm) | | ••• | | |
| Weight (kg) | | | | |
| BMI (kg/m^2) | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will continue for all categories of ethnicity and race

Height, Weight and BMI will be assessed using the same descriptive statistics as Age

If any values are missing, then a "missing" row will be included in the table, as applicable

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.1.4

Lifestyle Details: Smoking History and Alcohol Consumption

Summary Statistics: Safety Population

#### Sequence

| | | ABC <d> (N=X)</d> | BAC <d></d> | Overall (N=X) |
|---|---|---|---|---|
| Does the subject smoke? (1) | NO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PREVIOUSLY | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Alcohol Consumption (2) | NONE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | YES: NOT REGULARLY | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

- (1) Smoked or used e-cigarettes or nicotine replacement products in the last 12 months
- (2) Excessive alcohol consumption (>21 units/week in males and >14 units/week in females)
- 1 unit = 1/2 pint beer, 25 mL of 40% spirit, 1.5 to 2 units = 125 mL glass of wine depending on type

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Melinta Therapeutics Page x of y Protocol: ML-DEL-101-3727-1

TABLE 14.1.5

Extent of Exposure

Summary Statistics: Safety Analysis Set

| Regimen | Subjects Dosed (N=X) n (%) |
|---|---|
| 450 MG TAB FASTED | xx (xx.x) |
| 450 MG POS FASTED | xx (xx.x) |
| XXX MG POS <status> XXX MG POS <status></status></status> | xx (xx.x)<br>xx (xx.x) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

Arithmetic (1)

TABLE 14.2.1
Plasma Pharmacokinetic Concentrations: Delafloxacin <(units)>
Summary Statistics: <PK Analysis Set/PK Analysis Subset>

| | Arithmetic (1) | | | | | | | Geometric (2) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Regimen | Time Point | n | n# | Mean | SD | CV% | Median | Min | Max | Mean | SD | CV% |
| 450 MG TAB | PRE-DOSE | xx | xx | xx.xx | | xx.x | xx.xx | xx.x | | NC | NC | NC |
| FASTED | TIME POINT 1 | XX | XX | XX.XX | XX.XX | XX.X | xx.xx | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| (N=X) | TIME POINT 2 | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | TIME POINT 3 | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | | | | | | | ••• | ••• | | ••• | | ••• |
| | <all other="" points="" time=""></all> | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| 450 MG POS | PRE-DOSE | xx | XX | xx.xx | xx.xx | xx.x | xx.xx | xx.x | xx.x | NC | NC | NC |
| FASTED | TIME POINT 1 | XX | XX | xx.xx | xx.xx | XX.X | xx.xx | xx.x | XX.X | xx.xx | xx.xx | xx.x |
| (N=X) | TIME POINT 2 | XX | XX | XX.XX | xx.xx | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | xx.x |
| (14-25) | | | | | | | | | | | | |
| | TIME POINT 3 | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | ••• | | | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| | <all other="" points="" time=""></all> | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | | | ••• | | | | | | | | ••• | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> n# indicates the number of subjects with a BLQ value recorded at the time point indicated

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Geometric (2)

Programming note: This table will be continued for all time points Programming note: This table will be continued for all regimens

<sup>(1)</sup> For arithmetic summary statistics, concentration values reported as BLQ have been set to zero

<sup>(2)</sup> For calculation of geometric summary statistics, values reported as BLQ have been set to  $\frac{1}{2}$  × LLOQ, except for pre-dose values which will not be summarised. The LLOQ value was <value, units>

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.2.2

Plasma Pharmacokinetic Parameters: Delafloxacin

Summary Statistics: <PK Analysis Set/PK Analysis Subset>

| Regimen | Statistic | Parameter 1 (units) | Parameter 2 (units) | Parameter 3 (units) | All Other PK Parameters (units) |
|---|---|---|---|---|---|
| 450 MG TAB | n | XX | XX | XX | <br>xx |
| FASTED | Mean | xx.xx | XX.XX | XX.XX | <br>XX.XX |
| (N=X) | SD | XX.XX | XX.XX | XX.XX | <br>XX.XX |
| , , | CV% | XX.X | XX.X | XX.X | <br>XX.X |
| | Median | xx.xx | XX.XX | XX.XX | <br>XX.XX |
| | Min | XX.X | XX.X | XX.X | <br>XX.X |
| | Max | XX.X | XX.X | xx.x | <br>XX.X |
| | Geometric Mean | xx.xx | XX.XX | XX.XX | <br>xx.xx |
| | Geometric SD | XX.XX | XX.XX | XX.XX | <br>xx.xx |
| | Geometric CV% | XX.X | XX.X | XX.X | <br>XX.X |
| 450 MG POS<br>FASTED<br>(N=X) | | | | | <br> |
| | | | | ••• | <br> |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> For concentration parameters, BLQ values will be set to 0 for arithmetic statistics and to ½ × LLOQ for geometric statistics The LLOQ value was <value, units>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for all time points

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.2.3.1

Plasma Pharmacokinetic Parameters: Delafloxacin

450 MG POS

Statistical Analysis Results - Assessment of Relative Bioavailability: <PK Analysis Set/PK Analysis Subset>

450 MG TAB

| | | FASTED<br>(N=XX) | | FASTED<br>(N=XX) | | |
|---|---|---|---|---|---|---|
| Parameter | n | Adj Geo<br>Mean<br>(1) | n | Adj Geo<br>Mean<br>(1) | Ratio (%) | 90% CI<br>(3) |
| Cmax (units) | xx | xx.xx | xx | xx.xx | xx.xx | (xx.xx, xx.xx) |
| AUC(0-last) (units) | xx | xx.xx | xx | xx.xx | xx.xx | (xx.xx, xx.xx) |
| AUC(0-inf) (units) | XX | xx.xx | xx | xx.xx | xx.xx | (xx.xx, xx.xx) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Results obtained from mixed effects model of natural log transformed PK parameters including terms for regimen, period and sequence fitted as fixed effects and subject nested within sequence fitted as a random effect

(1) Adj geo mean = adjusted geometric mean from model (2) Ratio of adj geo means with comparison presented as test/reference (3) CI = confidence interval for ratio of adj geo means

PROGRAM PATH: X:\~\OSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.2.3.2

Plasma Pharmacokinetic Parameters: Delafloxacin

Statistical Analysis Results - Fixed Effects for Assessment of Relative Bioavailability: <PK Analysis Set/PK Analysis Subset>

| Parameter | Effect (1) | df (2) | F-Statistic (3) | p-value (4) |
|---------------------|------------|--------|-----------------|-------------|
| Cmax (units) | REGIMEN | xx,xx | x.xx | 0.xxx |
| , , | PERIOD | xx,xx | x.xx | 0.xxx |
| | SEQUENCE | xx,xx | x.xx | 0.xxx |
| AUC(0-last) (units) | REGIMEN | xx,xx | x.xx | 0.xxx |
| | PERIOD | xx,xx | x.xx | 0.xxx |
| | SEQUENCE | xx,xx | X.XX | 0.xxx |
| AUC(0-inf) (units) | REGIMEN | xx,xx | x.xx | 0.xxx |
| | PERIOD | xx,xx | x.xx | 0.xxx |
| | SEQUENCE | xx,xx | X.XX | 0.xxx |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Results obtained from mixed effects model of natural log transformed PK parameters including terms for regimen, period and sequence fitted as fixed effects and subject nested within sequence fitted as a random effect
(1) Fixed effects from the model (2) degrees of freedom for the fixed effects (3) F-statistic from the model for the relevant fixed effect (4) p-value for the relevant fixed effect

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.2.3.3

Plasma Pharmacokinetic Parameters: Delafloxacin

XXX MG POS

Statistical Analysis Results - Assessment of Food Effect: <PK Analysis Set/PK Analysis Subset>

XXX MG POS

| | < | STATUS><br>(N=XX) | | STATUS><br>(N=XX) | | |
|---|---|---|---|---|---|---|
| Parameter | n | Adj Geo<br>Mean<br>(1) | n | Adj Geo<br>Mean<br>(1) | Ratio (%) | 90% CI<br>(3) |
| Cmax (units) | xx | xx.xx | xx | xx.xx | xx.xx | (xx.xx, xx.xx) |
| AUC(0-last) (units) | XX | xx.xx | xx | xx.xx | xx.xx | (xx.xx, xx.xx) |
| AUC(0-inf) (units) | xx | xx.xx | xx | xx.xx | xx.xx | (xx.xx, xx.xx) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Results obtained from mixed effects model of natural log transformed PK parameters including terms for regimen, period and sequence fitted as fixed effects and subject nested within sequence fitted as a random effect
(1) Fixed effects from the model (2) degrees of freedom for the fixed effects (3) F-statistic from the model for the relevant fixed effect (4) p-value for the relevant fixed effect

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: a similar table will be produced for assessment of dose proportionality on dose corrected pk parameters if appliable, i.e. Table [14.2.3.4]

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.2.4 Taste/Palatability Assessments Taste/Palatability Analysis Set

<Overall Acceptability/Taste Attribute>

| Statistic | 450 MG POS<br>FASTED(N=XX) | XXX MG POS<br><status><br/>(N=XX)</status> | XXX MG POS<br><status><br/>(N=XX)</status> |
|---|---|---|---|
| n | xx | xx | xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | xx.x |
| GRADE 1 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 2 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 3 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 4 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 5 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 6 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 7 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 8 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 9 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Key for grade: 1 = Dislike extremely, 2 = Dislike very much, 3 = Dislike moderately, 4 = Dislike slightly, 5 = Neither like nor dislike, 6 = Like slightly, 7 = Like moderately, 8 = Like very much, 9 = Like extremely

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: Programming note: This table will be continued for all regimens A separate page will be used for each taste aspect and for overall acceptability with the relevant subheading

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.3.1

Overall Summary of Treatment-Emergent Adverse Events Summary Statistics: Safety Analysis Set

| | 450 MG TAB<br>FASTED<br>(N=X) | | 450 MG POS<br>FASTED<br>(N=X) | | XXX MG POS<br><status><br/>(N=X)</status> | | XXX MG POS<br><status><br/>(N=X)</status> | | Overall (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Event | n (%) | E | n (%) | E | n (%) | E | n (%) | E | n (%) | E |
| TEAE | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| Severe TEAE | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| ADR (1) | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| Serious TEAE | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| TEAE leading to subject/IMP withdrawa | l xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX |
| TEAE leading to death | xx (xx.x) | XX | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | xx |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> n is the number of subjects reporting at least one event. E = Total Number of Events

TEAEs are coded using MedDRA v27.0. (1) ADR is any AE where a causal relationship with the IMP is at least a reasonable possibility ie "possibly related" or "related"

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.3.2
Treatment-Emergent Adverse Events
By MedDRA System Organ Class and Preferred Term
Summary Statistics: Safety Analysis Set

| | FASTE | 450 MG TAB<br>FASTED<br>(N=X) | | 450 MG POS<br>FASTED<br>(N=X) | | XXX MG POS<br><status><br/>(N=X)</status> | | XXX MG POS<br><status><br/>(N=X)</status> | | Overall (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | n (%) | E | n (%) | E | n (%) | E | n (%) | E | n (%) | E |
| TEAEs | xx (xx.x) | XX | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | xx |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | XX | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| PREFERRED TERM 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| PREFERRED TERM 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| etc | | | | | | | | | | |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX |
| PREFERRED TERM 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| PREFERRED TERM 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| etc | | | | | | | | | ••• | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> n is the number of subjects reporting at least one event. E = Total Number of Events

TEAEs are coded using MedDRA v27.0 and are presented in descending order of frequency
Subjects experiencing more than one TEAE within a regimen are counted only once for number of subjects
but are counted more than once for number of events. Subjects experiencing more than one TEAE within a regimen are counted only once within each SOC and PT

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT

450 MG POS

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.3.3
Treatment-Emergent Adverse Events
By MedDRA System Organ Class, Preferred Term and Severity
Summary Statistics: Safety Analysis Set

| | | FASTED<br>(N=X) | | | | | |
|---|---|---|---|---|---|---|---|
| | Mild n(%) | | Severe<br>n(%) | Mild<br>n(%) | Moderate<br>n(%) | Severe<br>n(%) | |
| TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | <b></b> |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| etc | | | | | | | |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| etc | | | ••• | | | | |

450 MG TAB

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> TEAEs are coded using MedDRA v27.0 and are presented in descending order of frequency Counts are given for total number of subjects, not for events Counts of number of subjects are by maximum severity, ie subjects experiencing more than one TEAE within a regimen are counted only once within that regimen or each SOC and PT using the most severe episode

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT Programming note: This table will be continued for all regimens  $\frac{1}{2} \left( \frac{1}{2} \right) \left($ 

450 MG POS

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.3.4

Treatment-Emergent Adverse Events

By MedDRA System Organ Class, Preferred Term and Relationship to IMP

450 MG TAB

Summary Statistics: Safety Analysis Set

| | | FASTED<br>(N=X) | | | | | |
|---|---|---|---|---|---|---|---|
| | Unrelated n(%) | Possibly<br>Related<br>n(%) | Related n(%) | Unrelated n(%) | Possibly<br>Related<br>n(%) | Related n(%) | - |
| TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |
| etc | | | | | | | |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |
| etc | | | | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> TEAEs are coded using MedDRA v27.0 and are presented in descending order of frequency Counts are given for total number of subjects, not for events

Counts of number of subjects are by closest relationship, ie subjects experiencing more than one TEAE within a regimen are counted only once within that regimen or each SOC and PT using the most closely related event

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT Programming note: This table will be continued for all regimens  $\frac{1}{2} \left( \frac{1}{2} \right) \left($ 

Reporting and Analysis Plan ML-DEL-101-3727-1 (QSC300553) Final v1.0 24 Jun 2024 

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.3.5
Adverse Drug Reactions
By MedDRA System Organ Class and Preferred Term
Summary Statistics: Safety Analysis Set

| | | 450 MG<br>FASTE<br>(N=X | D | | 450 MG<br>FASTE<br>(N=X | |
|---|---|---|---|---|---|---|
| | | n (%) | E | | n(%) | E |
| ADRs (1) | xx | (xx.x) | xx | xx | (xx.x) | xx |
| SYSTEM ORGAN CLASS 1 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED TERM 1 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED TERM 2 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| etc | | | | | | |
| SYSTEM ORGAN CLASS 2 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED TERM 1 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED TERM 2 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| etc | | | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> n is the number of subjects reporting at least one event. E = Total Number of Events

TEAEs are coded using MedDRA v27.0 and are presented in descending order of frequency. <(1) An ADR is any AE where a causal relationship with the IMP is at least a reasonable possibility ie "possibly related" or "related">
Subjects experiencing more than one ADR within a regimen are counted only once for number of subjects but are counted more than once for number of events. Subjects experiencing more than one ADR within a regimen are counted only once within each SOC and PT

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for all regimens

Programming note: A similar table will be produced for Treatment-Emergent Serious Adverse Events, i.e. Table [14.3.6]

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.4.1 Haematology

Summary Statistics: Safety Analysis Set

<Parameter> (<units>) [ref range xxx-xxx (male), xxx-xxx (female)]

| | Time Point | | | F | Result | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Regimen | | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| 450 MG TAB | BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | |
| FASTED | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | XX.XX | xx.xx | XX.X | XX.X |
| (N=X) | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | XX.XX | xx.xx | XX.X | XX.X |
| | | | | | ••• | ••• | | | ••• | | | | |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| 450 MG POS | BASELINE | XX | xx.xx | xx.xx | XX.XX | xx.x | xx.x | | | | | | |
| FASTED | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| (N=X) | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | xx.xx | XX.X | XX.X |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | xx.xx | XX.X | XX.X |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral solution, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> BASELINE is defined as Day -1, Admission for Period 1 and Day 1, Pre-dose for Periods 2 to 4

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all haematology parameters and all time points

This table will be continued for all regimens

A similar table will be produced for Clinical Chemistry, i.e. Table [14.4.3]

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.4.1 Haematology

Summary Statistics: Safety Analysis Set

<Parameter> (<units>) [ref range xxx-xxx (male), xxx-xxx (female)]

| | Time Point | | | F | Result | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Regimen | | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| 450 MG TAB | BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | |
| FASTED | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| (N=X) | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| 450 MG POS | BASELINE | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | |
| FASTED | TIME POINT 1 | XX | xx.xx | XX.XX | XX.XX | XX.X | xx.x | XX | xx.xx | XX.XX | xx.xx | XX.X | XX.X |
| (N=X) | TIME POINT 2 | XX | xx.xx | XX.XX | xx.xx | XX.X | xx.x | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | | | | | | | | | | | ••• | | ••• |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> BASELINE is defined as Day -1, Admission for Period 1 and Day 1, Pre-dose for Periods 2 to 4

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all haematology parameters and all time points

This table will be continued for all regimens

A similar table will be produced for Clinical Chemistry, i.e. Table [14.4.3]

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.4.2 Haematology

Shift Analysis: Safety Analysis Set

<Parameter> (<units>) [ref range xxx-xxx (male), xxx-xxx (female)]

| | | | (N=X)<br>Baseline | | | (N=X)<br>Baseline | | |
|---|---|---|---|---|---|---|---|---|
| Time Point Assessment | N# | Below n(%) | Within Above Below n(%) n(%) N# n(%) | | Within<br>n(%) | Above<br>n(%) | | |
| TIME POINT 1 | xx | | | | xx | | | |
| Below | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Within | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Above | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TIME POINT 2 | XX | | | | xx | | | |
| Below | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Within | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Above | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |

450 MG TAB

FASTED

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> BASELINE is defined as Day -1, Admission for Period 1 and Day 1, Pre-dose for Periods 2 to 4

N# indicates the number of subjects with a baseline and a post baseline assessment at the time point indicated Below/within/above indicate the n(%)=number(%) of subjects with assessments below/within/above the normal reference range at

baseline

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

450 MG POS

FASTED

Programming note: This table will be continued for all haematology parameters and all time points Programming note: This table will be continued for all regimens

Reporting and Analysis Plan ML-DEL-101-3727-1 (QSC300553) Final v1.0 24 Jun 2024 

A similar table will be produced for Clinical Chemistry, i.e. Table [14.4.4]

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.5.1 Vital Signs

Summary Statistics: Safety Analysis Set

<Parameter> (<units>) [ref range xxx - xxx (age xx - xx), xxx - xxx (age > xx)]

| | Result | | | | | | | Change from<br>Baseline | | | | | | Substantial<br>Change (1) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max | DEC | NONE | INC |
| BASELINE | xx | | | xx.xx | xx.x | | | | | | | | | | |
| | XX | | | | XX.X | | XX | | | XX.XX | | | | XX | XX |
| | | | | | | | | | | | | | | | XX |
| TIME POINT 3 | XX | XX.XX | xx.xx | xx.xx | xx.x | XX.X | XX | xx.xx | XX.XX | xx.xx | XX.X | xx.x | XX | XX | XX |
| (711 other time points) | | | | | | | | | | | | | | | |
| <pre><aii other="" points="" time=""></aii></pre> | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | XX | XX.XX | xx.xx | xx.xx | xx.x | xx.x | XX | XX | XX |
| BASELINE | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | | | | |
| TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | xx.xx | XX.X | XX.X | XX | XX | XX |
| TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| TIME POINT 3 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | | | | ••• | | | | | | ••• | | | | | |
| <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | | ••• | | ••• | | | | ••• | | ••• | | | | | |
| | BASELINE TIME POINT 1 TIME POINT 2 TIME POINT 3 <all other="" points="" time=""> BASELINE TIME POINT 1 TIME POINT 2 TIME POINT 3 <all other="" points="" time=""></all></all> | BASELINE XX TIME POINT 1 XX TIME POINT 2 XX TIME POINT 3 XX <all other="" points="" time=""> XX BASELINE XX TIME POINT 1 XX TIME POINT 2 XX TIME POINT 3 XX <all other="" points="" time=""> XX</all></all> | BASELINE | ### Point N Mean SD ### BASELINE | ### Point N Mean SD Median ### BASELINE | Time Point N Mean SD Median Min | ### Point n Mean SD Median Min Max #### BASELINE | ### Point No Mean SD Median Min Max No No Median Min Max No No Median Min Max No No No Median Min Max No No No No No No No N | ### Point No. Mean SD Median Min Max No. Mean #### BASELINE XX | Result Baseline | Result | Result Baseline | Result Baseline | Result Baseline Ch. | Result Baseline Change |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> BASELINE is defined as Day 1, Pre-dose of the corresponding study period Substantial change is defined as: > ± 20 mmHg Systolic BP, > ± 10 mmHg Diastolic BP and > ± 15 bpm HR DEC: number of subjects with substantial decrease from baseline NONE: number of subjects with no substantial change from baseline, INC: number of subjects with substantial increase from baseline

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all vital signs parameters, which will follow the order given in the RAP text Programming note: This table will be continued for all regimens

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.5.2.1

ECGs

Summary Statistics: Safety Analysis Set

<Parameter> (<units>) [<ref range xxx - xxx (age xx - xx), xxx - xxx (age > xx)> / <ref range xxx - xxx (male), xxx-xxx (female)>]

| | | | | Re | esult | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Regimen | Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| 450 MG TAB | BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | |
| FASTED | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| (N=X) | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | xx.xx | XX.XX | XX.X | XX.X |
| | TIME POINT 3 | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| 450 MG POS | BASELINE | XX | XX.XX | xx.xx | xx.xx | XX.X | xx.x | | | | | | |
| FASTED | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | xx.xx | XX.XX | XX.X | XX.X |
| (N=X) | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIME POINT 3 | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | | | | ••• | | | | | | | | | |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | <b></b> | | | | | | | | | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> BASELINE is defined as Day 1, Pre-dose of the corresponding study period

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for all ECG parameters, which will follow the order given in the RAP text

Programming note: This table will be continued for all regimens

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

TABLE 14.5.2.2

ECGs

QTcF Categorical Data

Summary Statistics: Safety Analysis Set

| | | | QTcF (msec) | | | | | | | | | QTcF Increase<br>(msec) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | < | =450 | 4.5 | 51-480 | 48 | 31-500 | | >500 | | <=30 | 3 | 31-60 | | >60 |
| Regimen | Time Point | N# | n(%) | | n (%) | | n(%) | | n (%) | | n(%) | | n (%) | | | n(%) |
| 450 MG TAB | BASELINE | | XX | (xx.x) | XX | (xx.x) | xx | (xx.x) | XX | (xx.x) | | | | | | |
| FASTED | TIME POINT 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| (N=X) | TIME POINT 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| | TIME POINT 3 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| | <all other="" points="" time=""></all> | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| 450 MG POS | BASELINE | | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | XX | (xx.x) | | | | | | |
| FASTED | TIME POINT 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| (N=X) | TIME POINT 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| | TIME POINT 3 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| | <all other="" points="" time=""></all> | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> BASELINE is defined as Day 1, Pre-dose of the corresponding study period Categories for QTcF and QTcF increases are based on ICH E14 guidelines

N# is the number of subjects with a value at baseline and the relevant post-dose time point. It is the denominator for calculating the percentages of subjects, n indicates the number of subjects with observations at the given time point

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for all regimens
# 22 Mock Figures

Melinta Therapeutics 
Protocol: ML-DEL-101-3727-1

FIGURE 14.2.1.1
Plasma Pharmacokinetic Concentrations: Delafloxacin <(units)>
Linear/Linear Scale

Arithmetic Mean (± Arithmetic SD) Values: <PK Analysis Set/PK Analysis Subset>

All Fasted Regimens



Note: Data in the above graph are presented in Table [14.2.x.x]

Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Concentration values reported as <BLQ> have been set to 0 (LLOQ = x units). When all individual concentrations contributing to a mean become <BLQ>, the mean value for that time point will be presented as missing

PROGRAM PATH: Z:\~\QSCXXXXXX\~\TFLS\PRODUCTION\FIG-XX

DDMMMYYYY HH:MM

Programming note: Dummy data used. Axis lengths and labels will be updated as appropriate for this study

Programming note: This figure will be continued to show all Regimens

Programming note: Similar figure will be produced to show only the fed vs fasted comparison, i.e. Figure 14.2.1.3 and 14.2.1.4

Melinta Therapeutics

Protocol: ML-DEL-101-3727-1

FIGURE 14.2.1.2
Plasma Pharmacokinetic Concentrations: Delafloxacin <(units)>

 $\label{log10/Linear Scale} \begin{tabular}{ll} Log10/Linear Scale \\ Geometric Mean ($\times$/$\div Geometric SD) Values: $$<PK Analysis Set/PK Analysis Subset>$$$ 

All Fasted Regimens



Note: Data in the above graph are presented in Table [14.2.x.x]

Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Concentration values reported as <BLQ> have been set to ½ × LLOQ (LLOQ = x units). When all individual concentrations contributing to a mean become <BLQ>, the mean value for that time point will be presented as missing

Programming note: This figure will be continued to show all Regimens

Programming note: Similar figure will be produced to show only the fed vs fasted comparison, i.e. Figure 14.2.1.3 and 14.2.1.4

DDMMMYYYY HH:MM

Melinta Therapeutics
Page 1 of 2
Protocol: ML-DEL-101-3727-1

FIGURE 14.2.2.1

Plasma Pharmacokinetic Concentrations: Delafloxacin <(units)> Linear/Linear Scale

Spaghetti Plots of All Individual Values: <PK Analysis Set/PK Analysis Subset>

450 MG TAB FASTED



Note: Data in the above graph are presented in listing 16.2.x.x

Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Concentration values reported as <BLQ> have been set to 0 (LLOQ = x units), up until the point at which all of a subjects values become <BLQ>, then the values will be presented as missing

PROGRAM PATH: Z:\~\QSCXXXXXX\~\TFLS\PRODUCTION\FIG-SPAG
Programming note: Dummy data used. Axis lengths and labels will be updated as appropriate for this study

Each regimen will be presented on a seperate page

DDMMMYYYY HH:MM


Protocol: ML-DEL-101-3727-1

FIGURE 14.2.2.2 Plasma Pharmacokinetic Concentrations: Delafloxacin <(units)>Log10/Linear Scale

Spaghetti Plots of All Individual Values: <PK Analysis Set/PK Analysis Subset>

450 MG TAB FASTED



Note: Data in the above graph are presented in listing 16.2.x.x

Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Concentration values reported as <BLQ> have been set to ½ × LLOQ (LLOQ = x units), up until the point at which all of a subjects values become <BLQ>, then the values will be presented as missing

PROGRAM PATH: Z:\~\QSCXXXXXX\~\TFLS\PRODUCTION\FIG-SPAG

DDMMMYYYY HH:MM

Programming note: Dummy data used. Axis lengths and labels will be updated as appropriate for this study

Each regimen will be presented on a seperate page


Protocol: ML-DEL-101-3727-1

FIGURE 14.2.3.1

Plasma Pharmacokinetic Concentrations: Delafloxacin <(units)>
Linear/Linear Scale

Individual Values for Subject : <PK Analysis Set/PK Analysis Subset>



Note: Data in the above graph are presented in listing 16.2.x.x

Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Concentration values reported as <BLQ> have been set to 0 (LLOQ = x units), up until the point at which all of a treatments values become <BLQ>, then the values will be presented as missing

PROGRAM PATH: Z:\~\QSCXXXXXX\~\\TFLS\PRODUCTION\FIG-XX

DDMMMYYYY HH:MM

Programming note: Dummy data used. Axis lengths and labels will be updated as appropriate for this study

This figure will be continued to show all Regimens

This figure will be continued for all subjects


Protocol: ML-DEL-101-3727-1

FIGURE 14.2.3.2
Plasma Pharmacokinetic Concentrations: Delafloxacin <(units)>
Log10/Linear Scale

Individual Values for Subject < PK Analysis Set/PK Analysis Subset>



Note: Data in the above graph are presented in listing 16.2.x.x

Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Concentration values reported as <BLQ> have been set to ½ × LLOQ (LLOQ = x units), up until the point at which all of a treatments values become <BLQ>, then the values will be presented as missing

PROGRAM PATH: Z:\~\QSCXXXXXX\~\TFLS\PRODUCTION\FIG-XX

DDMMMYYYY HH:MM

Programming note: Dummy data used. Axis lengths and labels will be updated as appropriate for this study
This figure will be continued to show all Regimens
This figure will be continued for all subjects

Melinta Therapeutics 
Protocol: ML-DEL-101-3727-1

FIGURE 14.2.4.1

Plasma Pharmacokinetic Parameters: Delafloxacin

Adjusted Geometric Mean Ratio and 90% CIs: <PK Analysis Set/PK Analysis Subset>

450 MG TAB FASTED [test] vs 450 MG POS FASTED [reference]



Note: The data in this figure are presented in Table 14.2.X.X

Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>
Dashed lines represent the lower and upper limits of the bioequivalence assessment, i.e. 80.00% and 125.00%

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\FIG-XX

27MAY2024 11:25

Programming note: A similar figure will be produced for food effect analysis i.e., Figure [14.2.4.2]

# 23 Mock Listing

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

\_\_\_\_\_\_\_\_\_\_

LISTING 16.2.1

Subject Informed Consent and Completion/Withdrawal

Individual Values: All Enrolled Subjects

#### Informed Consent Form

| Subject<br>ID | Sex/<br>Age | Sequence | Date<br>Signed | Time<br>Signed | Version<br>Number | Did Subject<br>Complete<br>Study? | Completion/<br>Withdrawal<br>Date | Reason for<br>Withdrawal | Date of<br>Last Contact |
|---|---|---|---|---|---|---|---|---|---|
| XXX | M/35 | ABC <d></d> | DDMMMYYYY | HH:MM | XX | YES | DDMMMYYYY | | DDMMMYYYY |
| XXX | M/50 | ABC <d></d> | DDMMMYYYY | HH:MM | XX | NO | DDMMMYYYY | XXXX | DDMMMYYYY |
| XXX | M/50 | BAC <d></d> | DDMMMYYYY | HH:MM | XX | YES | DDMMMYYYY | | DDMMMYYYY |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: If no subjects withdraw, then 'Withdrawal Date' and 'Reason for Withdrawal' will not be presented

If re-consent is captured, then another Date/Time Signed and Version Number column will be added for re-consent

Melinta Therapeutics Page x of y Protocol: ML-DEL-101-3727-1

LISTING 16.2.2.1
Protocol Deviations

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Sequence | Period | Visit | Time<br>Point | Deviation<br>Date | Deviation Category/<br>Description of Deviation | Impact Assessment/ Impact Comment |
|---|---|---|---|---|---|---|---|---|
| XXX | M/35 | ABC <d></d> | | SCREENING | | DDMMMYYYY | XXXX/XXXX | MINOR |
| XXX | M/50 | ABC <d></d> | PERIOD 1 | DAY -1 | ADMISSION | DDMMMYYYY | XXXX/XXXX | MAJOR/XXXX |
| XXX | M/50 | BAC <d></d> | PERIOD 1 | DAY 1 | 3 Н | DDMMMYYYY | XXXX/XXXX | MINOR |
| | | <b></b> | | | | ••• | | *** |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: If no protocol deviations were reported, then a listing that states "NO PROTOCOL DEVIATIONS REPORTED" will be produced

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.2.2

Inclusion/Exclusion Criteria

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Sequence | All of Inclusion and<br>None of Exclusion Criteria | Criteria<br>Not Met | Criteria<br>Description |
|---|---|---|---|---|---|
| XXX | M/35 | ABC <d></d> | YES | | |
| XXX | M/50 | ABC <d></d> | YES | | |
| XXX | M/50 | BAC <d></d> | NO | EXCLUSION 2 | XXXX |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: If all subjects met all of the inclusion and none of the exclusion criteria, then a listing that states "ALL SUBJECTS MET THE ELIGIBILITY CRITERIA" will be produced

Melinta Therapeutics

Protocol: ML-DEL-101-3727-1

LISTING 16.2.3.1

Analysis Populations and Reasons for Exclusion Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Sequence | Population | Included in Population | Reason for Exclusion |
|---|---|---|---|---|---|
| XXX | М/35 | ABC <d></d> | SAFETY<br>PK<br>TASTE/PALATABILITY | YES<br>YES<br>YES | |
| XXX | M/50 | ABC <d></d> | SAFETY<br>PK<br>TASTE/PALATABILITY | YES<br>YES<br>YES | |
| XXX | M/50 | BAC <d></d> | SAFETY<br>PK<br>TASTE /PALATABILITY | NO<br>NO<br>NO | XXXX<br>XXXX<br>XXXX |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Page x of y

Programming note: A similar listing will be produced by treatment for

• Analysis Sets and Reasons for Exclusion, i.e. Listing [16.2.3.2]

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.1

Demographic and Baseline Characteristics Individual Values: All Enrolled Subjects

| Subjec<br>ID | t<br>Sequence | Age<br>(years) | Year of<br>Birth | Ethnicity | Race | Sex | Height (cm) | Weight<br>Screening<br>(kg) | Weight<br>Admission<br>(kg) | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | ABC <d></d> | XX | YYYY | XXXX | XXXX | MALE | XXX.X | XX.X | XX.X | XX.X |
| XXX | ABC <d></d> | XX | YYYY | XXXX | XXXX | MALE | XXX.X | XX.X | XX.X | XX.X |
| XXX | BAC <d></d> | XX | YYYY | XXXX | XXXX | MALE | XXX.X | XX.X | XX.X | XX.X |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.2

Lifestyle Details: Smoking History and Alcohol Consumption

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Sequence | Subject<br>Smoke | Date<br>Stopped | Subject<br>Drink<br>Alcohol | Units<br>per Week |
|---|---|---|---|---|---|---|
| XXX | M/35 | ABC <d></d> | PREVIOUSLY | DDMMMYYYY | YES | XX |
| XXX | M/50 | ABC <d></d> | NO | | YES | XX |
| XXX | M/50 | BAC <d></d> | NO | | NO | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

Melinta Therapeutics Page x of y Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.3

Medical/Surgical History

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Sequence | Category/<br>Description | System Organ Class/<br>Preferred Term | Date<br>of Onset | Date of<br>Resolution | Ongoing |
|---|---|---|---|---|---|---|---|
| XXX | M/35 | ABC <d></d> | NEUROLOGICAL/<br>XXXXXX | INFECTIONS AND INFESTATIONS/<br>MENINGITIS VIRAL | DDMMMYYYY | DDMMMYYYY | NO |
| XXX | M/50 | ABC <d></d> | REPRODUCTIVE/ | SURGICAL AND MEDICAL PROCEDURES/<br>VASECTOMY | DDMMMYYYY | | YES |
| | ••• | | | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Medical histories are coded using MedDRA v27.0

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.4

Prior and Concomitant Medication

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Sequence | M: Medication PT: Preferred Term ATC2: ATC Level 2 ATC4: ATC Level 4 I: Indication | R: Route<br>D: Dosage<br>U: Units<br>FRQ: Frequency | S: Start<br>E: End<br>O: Ongoing | P: Prior |
|---|---|---|---|---|---|---|
| XXX | M/35 | ABC <d></d> | M: XXXXXXXXXX PT: XXXXXXXXX ATC2: XXXXXXXXX ATC4: XXXXXXXX I: XXXXXXXX | R: XX<br>D: XXX<br>U: XX<br>FRQ: XXXXX XXXXX | S: DDMMMYYYY HH:M<br>E: DDMMMYYYY HH:M<br>O: NO | - " |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Medications are coded using the WHODrug Dictionary Global Drug Reference: 2024 Mar version (or a more recent version) Prior medications that start and stop prior to the first dose of IMP are flagged with a "#" symbol. Within this flagged group, medications that started after screening and stopped before dosing of IMP are also flagged using a "\*" symbol ATC = Anatomical Therapeutic Classification

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

Programming note: If no medications will be required from 14 days before IMP administration until discharge, then a listing that states "NO SUBJECTS REPORTED ANY PRIOR AND/OR CONCOMITANT MEDICATION" will be produced

DDMMMYYYY HH:MM

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.5 Urine Drug Screen

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Visit | Regimen | Date | Time | Parameter 1 | All Urine<br>Drug Parameters |
|---|---|---|---|---|---|---|---|
| XXX | M/35 | SCREENING | | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 1 DAY -1 | 450 MG TAB | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 2 DAY -1 | 450 MG POS | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 3 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 4 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| XXX | M/50 | SCREENING | | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 1 DAY -1 | 450 MG TAB | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 2 DAY -1 | 450 MG POS | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 3 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |
| | | PERIOD 4 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

Programming note: This listing will be continued for all urine drug parameters

DDMMMYYYY HH:MM

Melinta Therapeutics Page x of y Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.6

Alcohol and Carbon Monoxide Breath Test Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Visit | Regimen | Sample<br>Date | Alcohol<br>Breath Test | Carbon<br>Monoxide<br>Breath Test (ppm) |
|---|---|---|---|---|---|---|
| XXX | M/35 | SCREENING | | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 1 DAY -1 | 450 MG TAB | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 2 DAY -1 | 450 MG POS | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 3 DAY -1 | XXX MG POS | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 4 DAY -1 | XXX MG POS | DDMMMYYYY | NEGATIVE | XX |
| XXX | M/50 | SCREENING | | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 1 DAY -1 | 450 MG TAB | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 2 DAY -1 | 450 MG POS | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 3 DAY -1 | XXX MG POS | DDMMMYYYY | NEGATIVE | XX |
| | | PERIOD 4 DAY -1 | XXX MG POS | DDMMMYYYY | NEGATIVE | XX |
| | | | | <b></b> | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.7

Virology

Individual Values: All Enrolled Subjects

| Sample | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Sex/<br>Age | Sequence | Visit | Date | Time | Hepatitis B<br>Surface Antigen | Hepatitis C<br>Antibody | HIV Antibody |
| XXX | M/35 | ABC <d></d> | SCREENING | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE | NEGATIVE |
| XXX | M/50 | ABC <d></d> | SCREENING | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE | NEGATIVE |
| XXX | M/50 | BAC <d></d> | SCREENING | DDMMMYYYY | HH:MM | NEGATIVE | NEGATIVE | NEGATIVE |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

Melinta Therapeutics
Protocol: ML-DEL-101-3727-1

Page x of y

LISTING 16.2.4.8

Serum and Urine Pregnancy Test

Individual Values: All Enrolled Female Subjects

| | | | | Sample | | | |
|---|---|---|---|---|---|---|---|
| Subject<br>ID | Sex/<br>Age | Visit | Regimen | Date | Time | Test | Result |
| XXX | F/48 | SCREENING | | DDMMMYYYY | HH:MM | SERUM | NEGATIVE |
| | | PERIOD 1 DAY -1 | 450 MG TAB | DDMMMYYYY | HH:MM | URINE | NEGATIVE |
| | | PERIOD 2 DAY -1 | 450 MG POS | DDMMMYYYY | HH:MM | URINE | NEGATIVE |
| | | PERIOD 3 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | URINE | NEGATIVE |
| | | PERIOD 4 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | URINE | NEGATIVE |
| XXX | F/50 | SCREENING | | DDMMMYYYY | HH:MM | SERUM | NEGATIVE |
| | | PERIOD 1 DAY -1 | 450 MG TAB | DDMMMYYYY | HH:MM | URINE | NEGATIVE |
| | | PERIOD 2 DAY -1 | 450 MG POS | DDMMMYYYY | HH:MM | URINE | NEGATIVE |
| | | PERIOD 3 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | URINE | NEGATIVE |
| | | PERIOD 4 DAY -1 | XXX MG POS | DDMMMYYYY | HH:MM | URINE | NEGATIVE |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Melinta Therapeutics Page x of y Protocol: ML-DEL-101-3727-1

LISTING 16.2.4.9

Follicle Stimulating Hormone

Individual Values: All Enrolled Post-Menopausal Female Subjects

| 0-1-1 | Sex/ | | | Sampl | .e | DOU Analossia | |
|---|---|---|---|---|---|---|---|
| Subject<br>ID | Age | Sequence | Visit | Date | Time | FSH Analysis<br>Value (IU/L) | Reference Range |
| XXX | F/48 | ABC <d></d> | SCREENING | DDMMMYYYY | HH:MM | xxx.x | xxx.x - xxx.x |
| XXX | F/50 | ABC <d></d> | SCREENING | DDMMMYYYY | HH:MM | xxx.x | xxx.x - xxx.x |
| XXX | F/59 | BAC <d></d> | SCREENING | DDMMMYYYY | HH:MM | xxx.x | xxx.x - xxx.x |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

Melinta Therapeutics
Protocol: ML-DEL-101-3727-1

LISTING 16.2.5.1.1 Dosing Details

Individual Values: All Enrolled Subjects

| | | | | Do | sing | | | |
|---|---|---|---|---|---|---|---|---|
| Subject | Sex/ | | | | | Dose | Dose | Dose |
| ID | Age | Period | Regimen | Date | Time | Route | Form | Frequency |
| XXX | M/35 | PERIOD 1 | 450 MG TAB | DDMMMYYYY | нн:мм | xxx | XXXX | XXXX |
| | | PERIOD 2 | 450 MG POS | DDMMMYYYY | HH:MM | XXX | XXXX | XXXX |
| | | PERIOD 3 | XXX MG POS | DDMMMYYYY | HH:MM | XXX | XXXX | XXXX |
| | | <period 4=""></period> | XXX MG POS | DDMMMYYYY | HH:MM | XXX | XXXX | XXXX |
| XXX | M/50 | PERIOD 1 | 450 MG TAB | DDMMMYYYY | HH:MM | xxx | XXXX | XXXX |
| | | PERIOD 2 | 450 MG POS | DDMMMYYYY | HH:MM | XXX | XXXX | XXXX |
| | | PERIOD 3 | XXX MG POS | DDMMMYYYY | HH:MM | XXX | XXXX | XXXX |
| | | <period 4=""></period> | XXX MG POS | DDMMMYYYY | HH:MM | XXX | XXXX | XXXX |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.5.1.2

Meal Details for Fed Dosing

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Visit | Regimen | Meal<br>Description | Date | Start<br>Time | End<br>Time | Percent consumed (%) | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXX | M/35 | PERIOD 3 DAY 1<br>PERIOD 4 DAY 1 | XXX MG POS<br>XXX MG POS | XXXX | DDMMMYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM | HH:MM<br>HH:MM | XX - XX<br>XX - XX | XXXX XXXX |
| XXX | M/50 | PERIOD 3 DAY 1<br>PERIOD 4 DAY 1 | XXX MG POS<br>XXX MG POS | XXXX<br>XXXX | DDMMMYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM | HH:MM<br>HH:MM | XX - XX | XXXX XXXX |
| | | | | | | ••• | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.5.2

Blood Sample Collection Details for Pharmacokinetic Analysis and Plasma Pharmacokinetic Concentrations: Delafloxacin Individual Values: All Enrolled Subjects

| | | | | | | Sam | ple | | Parent | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Sex/ | | | | Time | | | Actual Time | Concentration | n | .Sample |
| ID | Age | Period | Regimen | Visit | Point | Date Time | | from Dose (h) | ( <units>)</units> | | Comments |
| XXX | M/35 | PERIOD 1 | 450 MG TAB | FDAY 1 | PRE-DOSE | DDMMMYYYY | HH:MM | XX.XX | BLO | | XXXX XXXX |
| | | | | | 0.5 H | DDMMMYYYY | HH:MM | XX.XX # | xx.x | | XXXX XXXX |
| | | | | | 1 H | DDMMMYYYY | HH:MM | XX.XX | XX.X | | XXXX XXXX |
| | | | | | 1.5 H | DDMMMYYYY | HH:MM | XX.XX | XX.X | | XXXX XXXX |
| | | | | | | | ••• | | | ••• | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> '#' indicates sample outside of scheduled time window.

BLQ = Below Limit of Quantification. Lower Limit of Quantification (LLOQ): XX ng/mL

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: Any exclusion from summary statistics due to non-evaluable profiles or timepoint will be shown by further footnotes and flagging

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.6.1

Plasma Pharmacokinetic Parameters: Delafloxacin Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Period | Regimen | PK Parameter 1 (units) | All<br>PK Parameters |
|---|---|---|---|---|---|
| XXX | M/35 | PERIOD 1 | 450 MG TAB | XXXX a d | XXXX |
| | , | PERIOD 2 | 450 MG POS | XXXX | XXXX |
| | | PERIOD 3 | XXX MG POS | XXXX | XXXX |
| | | <period 4=""></period> | XXX MG POS | XXXX | XXXX |
| XXX | M/50 | PERIOD 1 | 450 MG TAB | XXXX | XXXX |
| | | PERIOD 2 | 450 MG POS | XXXX c | XXXX a |
| | | PERIOD 3 | XXX MG POS | XXXX | XXXX |
| | | <period 4=""></period> | XXX MG POS | XXXX | XXXX |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Flags: a = Rsq of regression was <0.9, b = Period used for regression analysis was less than 2-fold the calculated half-life, c = Extrapolated portion of AUC(0-inf)>20%, d = Insufficient post-Cmax data points for estimation of lambda-z, e = Entire profile BLQ, no PK parameters could be calculated

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX DDMMMYYYY HH:MM

Programming note: Flags may be updated for emerging data

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.6.2 Taste Assessments

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Period | Regimen | Overall | Smell | Sweetness |
|---|---|---|---|---|---|---|
| XXX | M/35 | PERIOD 2<br>PERIOD 3 | 450 MG POS<br>XXX MG POS | XX<br>XX | XX<br>XX | XX<br>XX |
| | | | | ••• | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Key for grade: 1 = Dislike extremely, 2 = Dislike very much, 3 = Dislike moderately, 4 = Dislike slightly, 5 = Neither like nor dislike, 6 = Like slightly, 7 = Like moderately, 8 = Like very much, 9 = Like extremely, ND = not detectable

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.7.1

Pre-dose Adverse Events

Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | AE<br>No | System Organ Class/<br>Preferred Term/<br>Reported Term | Onset Date Time [Day (1)]/ End Date Time [Day (2)]/ Outcome [Duration (3)] | Serious/<br>Severity/<br>Relationship/<br>Cause if Not Related | Action<br>Taken |
|---|---|---|---|---|---|---|
| XXX | M/35 | XX | GASTROINTESTINAL DISORDERS/<br>ABDOMINAL PAIN/<br>ABDOMINAL ACHE (MILD) | DDMMMYYYY HH: MM [Day X]/<br>DDMMMYYYY HH: MM [Day X]/<br>RECOVERED/RESOLVED [X Days] | NO/<br>MILD/<br>NOT RELATED/<br>FOOD RELATED | NA |
| | | XX | | | | |
| | | | | | | ••• |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> AEs are coded using MedDRA v27.0

- (1) Study Day = Start date of AE Date of dose of IMP in study
- (2) Study Day = End date of AE Date of dose of IMP in study (+1 day if end date is on or post dose of IMP)
- (3) Duration (hours) = End date/time of AE Start date/time of AE

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: For (1) and (2), when the AE date is equal to or later than the IMP date then +1 day If AE is not resolved (2) and (3) will be missing

If no subjects experienced any pre-dose adverse events, then a listing that states

"NO SUBJECTS REPORTED ANY PRE-DOSE ADVERSE EVENTS" will be produced

"NO ADVERSE EVENTS RECORDED" will be specified for subjects with no pre-dose adverse events

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.7.2

All Treatment-Emergent Adverse Events Individual Values: All Enrolled Subjects

| Subject<br>ID | Sex/<br>Age | Period | Regimen | | System Organ Class/<br>Preferred Term/<br>Reported Term | Dose Date Time/ Onset Date Time [Day (1)]/ End Date Time [Day (2)]/ Outcome [Duration (3)] | Serious/<br>Severity/<br>Relationship/<br>Cause if<br>Not Related | Action<br>Taken |
|---|---|---|---|---|---|---|---|---|
| XXX | M/35 | PERIOD 1 | 450 MG TAB<br>FASTED | XX | GASTROINTESTINAL DISORDERS/<br>ABDOMINAL PAIN/<br>ABDOMINAL ACHE (MILD) | DDMMMYYYY HH: MM/<br>DDMMMYYYY HH: MM [Day X]/<br>DDMMMYYYY HH: MM [Day X]/<br>RECOVERED/RESOLVED [X Days] | NO/<br>MILD/<br>NOT RELATED/<br>FOOD RELATED | NA |
| | | PERIOD 2 | 450 MG POS<br>FASTED | XX | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> AEs are coded using MedDRA v27.0

- (1) Study Day = Start date of AE Date of dose of IMP +1 day
- (2) Study Day = End date of AE Date of dose of IMP +1 day
- (3) Duration (hours) = End date/time of AE Start date/time of AE

PROGRAM PATH: X:\~\OSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: For (1) and (2), the AE date is equal to or later than the IMP date, therefore +1 day

If AE is not resolved (2) and (3) will be missing

A similar listing will be produced for Serious Adverse Events, i.e. Listing [16.2.7.3] If no subjects experienced any treatment-emergent adverse events, then this listing will state "NO SUBJECTS REPORTED ANY TREATMENT-EMERGENT ADVERSE EVENTS". If no subjects experienced any

serious adverse events, then Listing [16.2.7.3] will state "NO SUBJECTS REPORTED ANY SERIOUS ADVERSE EVENTS"

"NO ADVERSE EVENTS RECORDED" will be specified for subjects with no adverse events

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.8.1

Blood Sample Collection Details for Laboratory Analysis

Individual Values: All Enrolled Subjects

| | | | | | | San | mple | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Sex/ | | | | Time | | | Samples | |
| ID | Age | Period | Regimen | Visit | Point | Date | Time | Obtained | Comments |
| XXX | M/35 | | | SCREENING | | DDMMMYYYY | HH:MM | AB | XXXX |
| | | PERIOD 1 | 450 MG TAB | DAY -1 | ADMISSION | DDMMMYYYY | HH:MM | AB | XXXX |
| | | | FASTED | DAY 1 | 2 H | DDMMMYYYY | HH:MM | AB | XXXX |
| | | PERIOD 2 | 450 MG POS | DAY -1 | ADMISSION | DDMMMYYYY | HH:MM | A | XXXX |
| | | | FASTED | DAY 1 | UNSCHEDULED # | DDMMMYYYY | HH:MM | A | XXXX |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> Sample Obtained: A = Clinical Chemistry, B = Haematology '#' indicates unscheduled observation

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: A similar listing will be produced for Urinalysis Sample Collection, i.e. Listing [16.2.8.6]

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.8.2 Haematology

Individual Values: All Enrolled Subjects

| Subject | Sex/ | | | Pariod | Period | | | Time | Sam | ple | (Refere | cameter<br>ence Range)<br>units) | Pai<br>(Refere | aematology<br>rameters<br>ence Range)<br>nits) * |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Age | Period | Regimen | Visit | Point | Date | Time | Value | Change | <br>Value | Change | | | |
| XXX | M/35 | PERIOD 1 | 450 MG TAB | SCREENING<br>DAY -1 | ADMISSION | DDMMMYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM | XX.X<br>XX.X H | | <br>XX.X<br>XX.X | | | | |
| | | PERIOD 2 | FASTED<br>450 MG POS<br>FASTED | <br>DAY 1<br>DAY 3 | <br>PRE-DOSE<br>48H | <br>DDMMMYYYY<br>DDMMMYYYY | <br>HH:MM<br>HH:MM | <br>XX.X H<br>XX.X L | <br>XX.X | <br><br>XX.X<br>XX.X | <br>XX.X | | | |
| | | | | | | <b></b> | | ••• | ••• | <br> | | | | |
| | | | | | | | | | ••• | <br> | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> H=Above normal reference range, L=Below normal reference range. <\* indicates a non-fasted, fasting sensitive, parameter> '#' indicates unscheduled observation
BASELINE is defined as Day -1, Admission for Period 1 and Day 1, Pre-dose for Periods 2 to 4

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: A similar listing will be produced for

• Clinical Chemistry, i.e. Listing [16.2.8.4]

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.8.3 Haematology

Individual Values Outside the Reference Range: All Enrolled Subjects

| Subject | Sex/ | | | | Time | Sample | | | | Reference |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Age | Period | Regimen | Visit | Point | Date | Time | Parameter | Result | Range |
| XXX | M/35 | PERIOD 1 | 450 MG TAB<br>FASTED | SCREENING<br>DAY -1<br> | ADMISSION | DDMMMYYYY<br>DDMMMYYYY<br> | НН:ММ<br>НН:ММ | XXXX (units)<br>XXXX (units)<br> | XX.X H<br>* XX.X L<br> | xx - xx<br>xx - xx |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> H=Above normal reference range, L=Below normal reference range. <\* indicates a non-fasted, fasting sensitive, parameter> '#' indicates unscheduled observation

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: Similar listings will be produced for

- Clinical Chemistry, i.e. Listing [16.2.8.5] and
- Urinalysis, i.e. Listing [16.2.8.8]

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.8.7 Urinalysis

Individual Values: All Enrolled Subjects

| | | | | | | Sam | ple | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Sex/ | | _ | | Time | | | | |
| ID | Age | Period | Regimen | Visit | Point | Date | Time | Parameter | |
| XXX | M/35 | | | SCREENING | | DDMMMYYYY | HH:MM | NEGATIVE | |
| | | PERIOD 1 | 450 MG TAB | DAY -1 | ADMISSION | DDMMMYYYY | HH:MM | NEGATIVE | ••• |
| | | | FASTED | DAY 1 | UNSCHEDULED # | DDMMMYYYY | HH:MM | NEGATIVE | |
| | | | | ••• | | | ••• | | |
| | | PERIOD 2 | 450 MG POS | DAY 1 | PRE-DOSE | DDMMMYYYY | HH:MM | NEGATIVE | |
| | | | FASTED | DAY 3 | 48 H | DDMMMYYYY | HH:MM | NEGATIVE | |
| | | | | ••• | | | ••• | ••• | ••• |
| | | | | ••• | ••• | | | ••• | ••• |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> All reference ranges are NEGATIVE/NORMAL unless otherwise specified

'#' indicates unscheduled observation

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.9.1.1 Vital Signs

Individual Values: All Enrolled Subjects

| | | | | | | Popu | ding | | ameter<br>nits) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Sex/ | | | Visit | Time | rea | arng | (unii cs) | | Clinical | |
| ID | Age | Period | Regimen | | Point | Date | Time | Value | Change | <br>Assessment | Findings |
| XXX | M/35 | | | SCREENING | | DDMMMYYYY | HH:MM | XXX | | <br>NORMAL | |
| | | PERIOD 1 | 450 MG TAB | DAY -1 | ADMISSION | DDMMMYYYY | HH:MM | XXX H | | <br>NORMAL | |
| | | | FASTED | DAY 1 | PRE-DOSE | DDMMMYYYY | HH:MM | XXX | XXX | <br>ABN, NCS | |
| | | | | | 1 H | DDMMMYYYY | HH:MM | XXX | XXX I | <br>ABN, NCS | |
| | | | | | 24 H | DDMMMYYYY | HH:MM | XXX | XXX | <br>NORMAL | |
| | | | | | | | | | | <br> | |
| | | PERIOD 2 | 450 MG POS | DAY -1 | ADMISSION | DDMMMYYYY | HH:MM | XXX | | <br>NORMAL | |
| | | | FASTED | DAY 1 | PRE-DOSE | DDMMMYYYY | HH:MM | XXX | XXX D | <br>NORMAL | |
| | | | | | 1 H | DDMMMYYYY | HH:MM | XXX | XXX | <br>ABN, NCS | |
| | | | | | 24 H | DDMMMYYYY | HH:MM | XXX | XXX | <br>ABN, CS | XXX |
| | | | | | ••• | | | ••• | | <br> | |
| | | | | | | | ••• | | ••• | <br> | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> H = Above normal reference range, L = Below normal reference range, I = Substantial Increase, D = Substantial Decrease Reference Ranges: Parameter 1 xx - xx <(units)> (xx-xx years), yy - yy <(units)> (yy-yy years), Parameter 2 xx - xx <(units)>, Parameter 3 xx - xx <(units)> (xx-xx years), yy - yy <(units)> (yy-yy years) Substantial change is defined as: > ± 20 mmHg Systolic BP, > ± 10 mmHg Diastolic BP and > ± 15 bpm HR BASELINE is defined as Day 1, Pre-dose of the corresponding study period. '#' indicates unscheduled observation ABN-NCS = Abnormal, not clinically significant.

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: This listing will be continued for all time points and subjects

The order of vital signs parameters is to be as per the order in the RAP text

Columns for 'Position' and 'Reading' will be included if samples are taken in multiple positions throughout the study and/or are taken in triplicate (lines for reading 1, 2, 3 and mean at each timepoint), respectively

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.9.1.2

Vital Signs

Individual Values Outside the Reference Range: All Enrolled Subjects

| | | | | | | Read | ding | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Sex/<br>Age | Period | Regimen | Visit | Time<br>Point | Date | Time | Parameter | Result | Reference<br>Range |
| XXX | M/35 | | | SCREENING | | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | xx - xx |
| | | PERIOD 1 | 450MG TAB | DAY -1 | ADMISSION | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | XX - XX |
| | | | FASTED | DAY 1 | PRE-DOSE | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | XX - XX |
| | | | | | 1 H | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | XX - XX |
| | | | | DAY 2 | 24 H | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | XX - XX |
| | | | | *** | *** | | ••• | | ••• | ••• |
| | | PERIOD 2 | 450 MG POS | DAY -1 | ADMISSION | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | XX - XX |
| | | | FASTED | DAY 1 | PRE-DOSE | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | XX - XX |
| | | | | | 1 H | DDMMMYYYY | HH:MM | XXXX (units) | XXXX H | XX - XX |
| | | | | DAY 2 | 24 H | DDMMMYYYY | HH:MM | XXXX (units) | XXXX L | XX - XX |
| | | | | ••• | ••• | | *** | | ••• | |
| ••• | ••• | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> H = Above normal reference range, L = Below normal reference range

Listing contains all data outside the normal reference range for all vital signs parameters at the relevant time points '#' indicates unscheduled observation

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: This listing will be continued for all data outside the reference range, for all relevant vital sign parameters and for all time points, as applicable. If no values were recorded outside of the reference range, then a listing that states 'NO VALUES OUTSIDE THE REFERENCE RANGE WERE RECORDED' will be produced

A similar listing will also be produced for

• ECGs (Values Outside the Reference Range), i.e. Listing [16.2.9.2.2] and

Melinta Therapeutics
Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.9.2.1

ECGs

Individual Values: All Enrolled Subjects

| | | | | | | Read | ing | Para | meter | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Sex/<br>Age | Period | Regimen | Visit | Time<br>Point | Date | Time | Value<br>(units) | Change<br>(units) | Rhythm | Interpretation |
| _ | | | | | | | | | | | |
| XXX | M/35 | PERIOD 1 | 450 MG TAB<br>FASTED | SCREENING<br>DAY -1<br>DAY 1 | ADMISSION<br>PRE-DOSE<br>1 H<br>24 H | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM | XXX H<br>XXX<br>XXX<br>XXX | XXX I | SINUS RHYTHM SINUS RHYTHM SINUS RHYTHM SINUS RHYTHM SINUS RHYTHM | NORMAL<br>NORMAL<br>NORMAL<br>NORMAL<br>NORMAL |
| XXX | | PERIOD 2 | 450 MG POS<br>FASTED | SCREENING DAY -1 DAY 1 DAY 2 | ADMISSION PRE-DOSE 1 H 24 H | DDMMMYYYY DDMMMYYYY DDMMMYYYY DDMMMYYYY DDMMMYYYY | HH: MM<br>HH: MM<br>HH: MM<br>HH: MM<br>HH: MM | XXX H XXX XXX XXX | XXX XXX SI XXX | SINUS RHYTHM SINUS RHYTHM SINUS RHYTHM SINUS RHYTHM SINUS RHYTHM SINUS RHYTHM INUS RHYTHM INUS RHYTHM | NORMAL NORMAL ABNORMAL, NCS, NORMAL ABNORMAL, CS, XXX |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status> H = Above normal reference range, L = Below normal reference range, I = Increase in QTcF from baseline 31-60 msec, SI = Substantial Increase in QTcF Reference Ranges: Parameter 1 xx - xx <(units)> (xx-xx years), yy - yy <(units)> (yy-yy years), Parameter 2 xx - xx <(units)>, Parameter 3 xx - xx <(units)> (xx-xx years), yy - yy <(units)> (yy-yy years) Substantial Increase in QTcF from baseline defined as >60 msec BASELINE is defined as Day 1, Pre-dose of the corresponding study period. '#' indicates unscheduled observation NCS = Not clinically significant. CS = Clinically significant

PROGRAM PATH: X:\~\OSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: This listing will be continued for all time points and subjects The order of ECG parameters is to be as per the order in the RAP text

Reporting and Analysis Plan ML-DEL-101-3727-1 (QSC300553) Final v1.0 24 Jun 2024 

Melinta Therapeutics Page x of y
Protocol: ML-DEL-101-3727-1

LISTING 16.2.9.3

Physical Examination Data

Individual Values: All Enrolled Subjects

#### Physical Examination

| Subject | Sex/ | | | | | JAdilliaci | 011 | Targeted/ | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Age | Period | Regimen | Visit | Date | Time | Performed | Planned | Body System | Result |
| XXX | M/35 | PERIOD 1 | 450 MG TAB<br>FASTED | SCREENING<br>DAY -1 | DDMMMYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM | XXX | XXX | ALL BODY SYSTEMS<br>MUSCULOSKELETAL | XXX |
| | | | ••• | | | ••• | | | | |

Note: Investigational Medicinal Product is delafloxacin, POS = powder for oral suspension, Regimen B, C and D with orange flavour Regimen Key: A = 450 mg tablet (reference) fasted, B = 450 mg POS fasted, C = xxx mg POS <status>, D = xxx mg POS <status>

PROGRAM PATH: X:\~\QSCXXXXXX\~\TFLS\PRODUCTION\LIS-XX

DDMMMYYYY HH:MM

Programming note: This listing will be continued for all time points and subjects

## **Appendix 1: Schedule of Assessments**

| Study Day | -28 | -1 | | 1<br>Times After Dosing (h) | | | | | | | | | | 2 | 3 | 6 ± 1 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | to -2 | | | | | | | | Tim | es Af | ter Do | sing ( | h) | | | | | | | FUP Phone Call |
| | S | Aª | Р | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 48 <sup>b</sup> | or Unscheduled<br>FUP Visit <sup>c</sup> |
| General Assessments | | | | | | | | | | | | | | | | | | | | |
| Informed Consent | Х | | | | | | | | | | | | | | | | | | | |
| Medical History | X | $X^d$ | | | | | | | | | | | | | | | | | | |
| Weight, Height and BMI | Х | Xe | | | | | | | | | | | | | | | | | | |
| Vein Assessment | Х | Xf | | | | | | | | | | | | | | | | | | |
| Drug Screen | Х | Х | | | | | | | | | | | | | | | | | | |
| Alcohol Breath Test | Х | Χ | | | | | | | | | | | | | | | | | | |
| Carbon Monoxide Breath Test | Х | Χ | | | | | | | | | | | | | | | | | | |
| Randomisation <sup>g</sup> | | | Χ | | | | | | | | | | | | | | | | | |
| IMP Administration | | | | Х | | | | | | | | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | | | | | | | | |
| Physical Examination | Х | | | | | | | | | | | | | | | | | | | |
| Targeted (symptom driven) Physical<br>Examination <sup>h</sup> | | X <sup>f</sup> | Xi | | | | | | | | | | | | | | | х | | Х |
| Clinical Laboratory Tests <sup>j</sup> | Х | Xf | Xi | | | | | | | | | | | | | | | | Х | X |
| Urinalysis | Х | X <sup>f</sup> | Χ <sup>i</sup> | | | | | | | | | | | | | | | | Х | |
| Serum Pregnancy Test <sup>k</sup> | Х | | | | | | | | | | | | | | | | | | | |
| Urine Pregnancy Test <sup>k</sup> | | Χ | | | | | | | | | | | | | | | | | Х | X |
| Single 12-Lead ECGs | Х | Χ | Χ | | | Х | | | | | | | | | | | | Х | Х | X |
| Vital Signs <sup>l</sup> | Х | Χ | Χ | | | Х | | | | | | | | | | | | Х | Х | X |
| Adverse Events | < | | | | | | | | | | X | | | | | | | | | > |
| Prior and Concomitant Medication | < | | | | | | | | | | X | | | | | | | | | > |
| PK Assessments | | | | | | | | | | | | | | | | | | | | |
| Plasma Samples for Delafloxacin | | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Taste/Palatability Assessments | | | | | | | | | | | | | | | | | | | | |
| Taste/Palatability Questionnaire <sup>m</sup> | | | | Х | | | | | | | | | | | | | | | | |
| $\Delta$ = admission FLIP = follow-up P = | d | 200 | = 00r | oning | | | | | | | | | | | | | | | | |

A = admission, FUP = follow-up, P = pre-dose, S = screening

If replacement subjects are required, they will undergo screening assessments as detailed above

All assessments/procedures to be completed for every period unless specified otherwise

<sup>&</sup>lt;sup>a</sup> Subjects will be admitted to the clinical unit in the morning on the day before dosing (Day -1) in Period 1, and in the evening on the day before dosing (Day -1) in Period 3 and optional Period 4. Subjects will remain resident in the clinical unit between Periods 1 and 2; therefore, no admission procedures will be conducted for Period 2

- <sup>b</sup> Discharge from the clinical unit (Periods 2 to 4 only). There will be a minimum washout of 4 days between dosing in Periods 1 and 2. In the event of early withdrawal, discharge assessments should be completed
- <sup>c</sup> A follow-up phone call will take place on Day 6 ± 1 of the final treatment period, to ensure the ongoing wellbeing of the subjects. If a subject reports any AEs that present a cause for concern, they will be required to attend the clinical unit for a (unscheduled) follow-up visit. Assessments may be performed at the unscheduled follow-up visit as indicated
- d Update only
- e Weight only
- f Period 1 only
- <sup>9</sup> Subjects will be randomised immediately prior to dosing in Period 1, for allocation of regimens across Periods 1 and 2
- h Targeted (symptom driven) physical examination of the relevant body system(s) as clinically indicated, as per the Investigator's judgement
- Periods 2 to 4 only
- <sup>1</sup> Haematology and clinical chemistry at each time point including virology and FSH (post-menopausal female subjects only) at screening
- <sup>k</sup> All female subjects
- <sup>1</sup> Blood pressure, heart rate, oral temperature and respiratory rate will be measured at each time point
- <sup>m</sup> The taste/palatability questionnaire will be started within 10 minutes of each delafloxacin Powder for Oral Suspension (i.e., test) regimen administration. See Appendix 2 for details of the taste/palatability questionnaire

#### **Appendix 2: Example Taste/Palatability Questionnaire** QSC300553 (ML-DEL-101-3727-1) Taste Questionnaire **Study Period:** Regimen: **Subject Number: Subject Initials:** Start time: (to be started within 10 minutes of dosing) Date: **Question 1** All aspects considered (smell, sweetness, bitterness, flavour, mouthfeel/texture, grittiness, and aftertaste), how would you rate your overall liking of this product: NOTE: Tick 1 box below in blue or black pen Dislike Dislike very Dislike Neither like nor Like Dislike slightly Like slightly Like very much Like extremely extremely much moderately dislike moderately Question 2

We want to know how much you like certain aspects of the product: smell, sweetness, bitterness, flavour, mouthfeel/texture, grittiness, and aftertaste. Please rate each test product independently of any previous taste questionnaires. NOTE: Tick 1 box in the row for each aspect

| | Dislike extremely | Dislike very much | Dislike<br>moderately | Dislike<br>slightly | Neither like nor dislike | Like slightly | Like<br>moderately | Like very<br>much | Like<br>extremely | Not<br>detectable |
|---|---|---|---|---|---|---|---|---|---|---|
| Smell | | | | | | | | | | |
| Sweetness | | | | | | | | | | |
| Bitterness | | | | | | | | | | |
| Flavour | | | | | | | | | | |
| Mouthfeel/texture | | | | | | | | | | |
| Grittiness | | | | | | | | | | |

# Aftertaste Entered into eCRF by (initials): Date: Confidential QC checked by (initials): Date: